#### **TITLE**

# PHASE I - II STUDY OF PRONE ACCELERATED BREAST AND NODAL IMRT

**Coordinating Center:** New York University Cancer Institute

160 East 34<sup>th</sup> Street New York, NY 10016

\*Principal Investigator: Carmen Perez, M.D.

160 East 34<sup>th</sup> Street New York, NY 10016 Telephone: (212) 731-5003 Fax: (212) 731-5513

E-mail address: carmen.perez@nyumc.org

**Co-PI:** Silvia.C.Formenti, M.D.

160 East 34<sup>th</sup> street New York, NY – 10016 Telephone : 212-731-5003 *Fax: (212) 731-5513* 

E-mail address: silvia.formenti@nyumc.org

Co-Investigators:

Nelly Huppert, M.D. 160 East 34<sup>th</sup> Street New York, NY 10016 Telephone: (212) 731-5030 Fax: (212) 731-5512

E-mail address: nelly.huppert@nyumc.org

Joshua Silverman, M.D. 160 East 34<sup>th</sup> Street New York, NY 10016

Telephone: (212) 731-5880

Fax: (212) 731-5512

E-mail address: joshua.silverman2@nyumc.org

Brian Yeh, M.D. 160 East 34th Street

New York, NY 10016

Telephone: (212) 731-5044

Fax: (212) 731-5512

E-mail address:brian.yeh@nyumc.org

Linda Moy, M.D. 560 First Avenue New York, NY 10016

Telephone: (212) 731-5353 E-mail: Linda.Moy@nyumc.org

Adrienne Newburg, M.D. 550 First Avenue New York, NY 10016 Telephone: (212) 263-7300

E-mail: Adrienne.Newburg@nyumc.org

Barry Rosenstein, Ph.D. 1 Gustave L. Levy Place New York, NY 10029 Telephone: (212) 241 9408

Fax: (212) 996 8927

E-mail address: barry.rosenstein@mssm.edu

Naamit Gerber, M.D.

160 East 34th Street

New York, NY 10016

Telephone: (212) 731-5003

Fax: (212) 731-5512

E-mail address: Naamit.Gerber@nyumc.org

Olivier Maisonet, N.P. 160 East 34th Street New York, NY 10016 Telephone: (212) 731-5035

Fax: (212) 731-5512

E-mail address: Olivier. Maisonet@nyumc.org

Judith D. Goldberg, Sc.D. (Biostatistics) 650 First Avenue, KIP 5 534

New York NY 10016 Telephone: (212) 263 0314 Fax: (212) 263 8570

E-mail address: jd.goldberg@nyumc.org

# **TABLE OF CONTENTS**

| | | | Page |
|---|---|---|---|
| SC | HEM | A | 7 |
| LIS | ST OF | F ABBREVIATIONS AND DEFINITION OF TERMS | 8 |
| 1. | OR. | JECTIVES | 9 |
| -• | 1.1 | Primary Objectives | |
| | 1.2 | Secondary Objectives | |
| 2. | BAG | CKGROUND | 9 |
| | 2.1 | NYU Research in Hypofractionated Whole Breast Radiotherapy | 9 |
| | 2.2 | NYU Experience on Accelerated Concomitant Boost Whole Breast: NYU 03 | |
| | 2.3 | Rationale for Prone Radiotherapy: NYU 05-181 | |
| | 2.4 | Rationale for Treating Axillary Level III and Supraclavicular Nodes | 12 |
| | 2.5 | Late Radiation Effects and Assessment of Risk | |
| | 2.6 | Dose Selection for Treating Breast and Nodal Stations | |
| | 2.7 | Quality of Life Assessment | |
| | 2.8 | Measuring the Late Toxicities of Breast and Nodal Radiation | 21 |
| 3 | PAT | FIENT SELECTION | 23 |
| | _ ~ ~ | | |
| | | PHORT A : INCLUDE PATIENTS WHO HAVE UNDERGONE SLNB UT COMPLETION ALND) | 23 |
| *** | 3.1 | Inclusion Criteria | |
| | 3.2 | Exclusion Criteria | |
| 4 | REC | GISTRATION PROCEDURES | 24 |
| - | 4.1 | General Guidelines | |
| | 4.2 | Registration Process | |
| 5 | TRI | EATMENT PLAN | 25 |
| | 5.1 | General Concomitant Medication and Supportive Care Guidelines | |
| | 5.2 | Duration of Therapy | |
| | 5.3 | Duration of Follow-up | |
| | 5.4 | Alternatives | |
| | 5.5 | Compensation | |
| 6 | SUF | RGERY | 25 |
| 7 | RA | DIOTHERAPY SPECIFICATIONS | 26 |
| | 7.1 | Treatment Planning using Hybrid IMRT Technique | |
| | 7.2 | Dose Specification | |
| | 73 | CT Simulation | 26 |

| | 7.4 | Target Delineation | 27 |
|---|---|---|---|
| | 7.5 | Technical Factors | |
| | 7.6 | Portal Imaging | |
| 8 | DOS | E MODIFICATIONS AND STOPPING CRITERIA | |
| | 8.1 | Dose Modification | 29 |
| | 8.2 | Stopping Criteria | 29 |
| 9 | ADV | TERSE EVENTS: LIST AND REPORTING REQUIREMENTS | |
| | 9.1 | Adverse Events and Potential Risks List | |
| | 9.2 | Expedited Adverse Event Reporting | |
| | 9.3 | Routine Adverse Event Reporting Guidelines | 30 |
| 10 | COR | RRELATIVE/SPECIAL STUDIES | |
| | 10.1 | Blood Collection for TGF-beta 1 Polymorphism Determination | |
| | 10.2 | Lymphocyte Isolation, DNA Extraction, PCR Amplification and DNA Sequencing | |
| | 10.3 | Test Method | |
| | 10.4 | Denaturing High Performance Liquid Chromatography (DHPLC) | |
| | 10.5 | Coding of Samples | 32 |
| 11 | INV | ESTIGATOR RESOURCES | 32 |
| | 11.1 | Qualifications | |
| | | Use of NYU Facilities | |
| | 11.3 | Conflict of Interest | 33 |
| 12 | STU | DY CALENDAR | 34 |
| 13 | DAT | 'A REPORTING / REGULATORY CONSIDERATIONS | 34 |
| | 13.1 | Monitoring Plan | 34 |
| | 13.2 | Stopping Rules (for the individual patient and for the study as a whole) | 35 |
| | 13.3 | Data Management | 35 |
| | 13.4 | Confidentiality | 35 |
| 14 | STA | TISTICAL CONSIDERATIONS | 36 |
| | 14.1 | Endpoints/Objectives: | |
| | 14.2 | Statistical Considerations, Sample Size and Interim Analysis Plans | 36 |
| | 14.3 | Statistical Analysis | 36 |
| | 14.4 | Accrual estimates | 37 |
| | 14.5 | Sample Size Considerations/Interim Analysis | 37 |
| RE] | FERE | NCES | 39 |
| API | PEND | IX 1 – COMMON TOXICITY CRITERIA | 43 |
| | | IX 2 – TOXICITY TRACKING FORM | |
| 4 <b>31</b> 1 | | 17 2 1 0/MOITT TRACKING FORM | - |

| APPENDIX 3 – QUALITY OF LIFE QUEST PROTOCOL SYNOPSIS | TIONNAIRES 46 |
|---|---|
| TITLE | Phase I - II Study of Prone Accelerated Breast and Nodal IMRT |
| STUDY PHASE | I - II |
| INDICATION | Stage II - III breast cancer (AJCC 2002) |
| PRIMARY OBJECTIVES | Feasibility, Acute toxicity |
| SECONDARY OBJECTIVES | Incidence of re-simulation supine, |
| | QOL (defined by RTOG-PRO), |
| | Late toxicity: e.g., fibrosis, telangiectasia, |
| | Local control: Time to Progression, |
| EXPLORATORY OBJECTIVES | Survival and evaluation of genetic determinants of breast fibrosis |
| HYPOTHESES | Prone IMRT to breast, level III and SCV nodes is feasible and well tolerated in a 3-week regimen |
| STUDY DESIGN | Prospective, single arm uncontrolled |
| PRIMARY ENDPOINTS | Acute, late effects, QOL-PRO |
| SAMPLE SIZE BY TREATMENT GROUP | 104 patients. Cohort A – 30 patients |
| SUMMARY OF SUBJECT ELIGIBILITY CRITERIA | Newly diagnosed breast cancer patients after segmental mastectomy, and axillary dissection of at least 8 lymph nodes. |
| INVESTIGATIONAL PRODUCTS DOSAGE AND ADMINISTRATION | N/A |
| CONTROL GROUP | N/A |

N/A

Phase I - II

STATISTICAL CONSIDERATIONS

**PROCEDURES** 

#### **SCHEMA**

# ELIGIBLE PATIENTS INFORMED CONSENT

Whole breast/chest wall, level 1- III (includes Cohort A) and SCV nodes IMRT at 2.7 Gy x 15 fractions

Total dose to the indexed breast = 40.50 Gy

Daily 0.5 Gy boost to the tumor bed (15 fractions)

Total dose to tumor bed = 48 Gy

All patients will be followed for toxicity and outcome (i.e., local and systemic recurrence, survival). In addition, patients will complete a Quality of Life (QOL) self-assessment at baseline, week 3, day 45-60 and 2-yr follow-ups.

#### LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

ADL Activities of daily living

AE Adverse event

ATM Ataxia Telangiectasia Mutated
BED Biologically Effective Dose
CBC Complete blood count
CI Confidence interval

Cone-Beam CT

CRF Case report/Record form

CTCAE Common Terminology Criteria for Adverse Events

CTV Clinical target volume
DCIS Ductal Carcinoma In Situ

DHPLC Denaturing High Performance Liquid Chromatography

DSMB Data Safety Monitoring Board

ECG Electrocardiogram

Gy Gray

**CBCT** 

Hgb Hemoglobin

IBV Ipsilateral Breast Volume

IMRT Intensity Modulated RadioTherapy

IRB Institutional Review Board

LENT/SOMA Late Effects Normal Tissues / Subjective, Objective, Management

criteria with Analytic laboratory and imaging procedures

LLN Lower limit of normal OS Overall survival

PCR Polymerase Chain Reaction

PCR-RFLP Polymerase Chain Reaction-Restriction Fragment Length Polymorphism

PD Progressive Disease PFS Progression free survival

PLT Platelet

PR Partial response

PTT Protein Truncation Test
PTV Planning Target Volume

QOL Quality of Life

RBV Residual Breast Volume
RIF Radiation-Induced Fibrosis

RR Response rate

RTOG Radiation Therapy Oncology Group

SAE Serious adverse event

SD Stable disease

SNP Single Nucleotide Polymorphism

SSCP Single-Strand Conformation Polymorphism

TGF-beta1 Transforming Growth Factor beta-1

TV Treatment Volume

#### 1. OBJECTIVES

#### 1.1 Primary Objectives

1.1.1 To evaluate feasibility of prone IMRT to breast, level III and supraclavicular nodes (physics and dosimetry parameters)

1.1.2 To estimate acute toxicity of prone IMRT to breast, level III and supraclavicular nodes

#### 1.2 Secondary Objectives

- 1.2.1 To estimate the incidence of re-simulation to improve dosimetry after initial prone set-up
- 1.2.2 To evaluate changes in QOL of patients assessed at baseline and after treatment
- 1.2.3 To estimate incidence of late radiation toxicity (e.g., lymphedema, fibrosis and telangiectasia) and to examine genetic determinants of breast fibrosis

# 1.3 Exploratory Objectives

- 1.3.1 To estimate local recurrence rates
- 1.3.2 To estimate median Disease Free Survival (DFS)
- 1.3.3 To estimate median Time to Progression
- 1.3.4 To estimate median Overall Survival (OS)

#### 1.4 Cohort A Objectives

1.4.1 To explore feasibility of treating in the prone position a comprehensive nodal volume, that includes axillary nodal levels I and II in addition to the fields already treated per this protocol (i.e., axillary nodal levels III, supraclavicular fossa and breast or chest wall tangents, depending on whether the patient has undergone segmental mastectomy or mastectomy, respectively)

#### 2. BACKGROUND

2.1 NYU Research in Hypofractionated Whole Breast Radiotherapy

A recent Cochrane Collaboration Intervention Review has addressed the effects of altered fractionation size on women with early breast cancer who have undergone breast conservation surgery (James Melissa, Lehman et al. 2008). Analysis of two prospective randomized trials that included 2644 women, selected based on tumor size less than five cm, negative pathological margin of excision and negative lymph nodes. No difference in clinical outcome was detected. The conclusion of the review is that the use of unconventional fractionation regimens (greater than 2 Gy per fraction) does not affect breast appearance or toxicity, and does not seem to affect local recurrence or five years survival rates.

Hypofractionation regimens enable shortening of the duration of therapy; the findings are quite relevant, since changing the standard recommendation of 30 fractions over six weeks to a 3week regimen could result in higher compliance and cost saving.

During the past eight years the Breast Cancer Radiotherapy Research team at NYU has conducted a series of consecutive studies to optimize the safe delivery of accelerated radiotherapy to partial and whole breast. As background for the proposed study that will test a novel technique to target the breast and level III/SCV nodes in the prone position for women with 1 - 5 involved nodes, a review of the whole breast radiation research studies conducted thus far is detailed below.

NYU Experience on Accelerated Concomitant Boost Whole Breast: NYU 03-30

Inspired by the hypo-fractionated Canadian trial (Whelan, MacKenzie et al. 2002) we developed a technique that utilizes IMRT to deliver accelerated prone whole breast radiotherapy with a concomitant boost to the tumor bed. The rationale for adding a boost to the tumor cavity derived from the results of a prospective randomized trial conducted by the EORTC (Bartelink, Horiot et al. 2001). A recent update of the trial demonstrated a 10-year cumulative incidence of local recurrence of 10.2% versus 6.2% for the no boost and the boost group respectively (p < 0.0001) (Bartelink, Horiot et al. 2007).

Patients with stage I or II breast cancer, excised by breast conserving surgery with negative margins, and either sentinel node biopsy or axillary dissection were eligible for study NYU 03-30. CT simulation was performed with the patient on a dedicated prone breast board, in the exact position used for treatment.

From September 2003 to August 2004, the planned accrual was completed, with 90 patients treated in the protocol (mean follow-up of 39 months, range 1 - 72 months). Median age was 58 years old (range 28 – 80 yo). Median tumor size was 13 mm (range 1 - 40 mm). Acute toxicity was generally mild and is summarized in Table 1 (RTOG score). Most common toxicity was radiation dermatitis, which tended to occur the week after completion of treatment.

| | Grade 1 | Grade2 | Grade 3 | Grade 4 |
|--------------|----------|---------|---------|---------|
| Dermatitis | 38 (42%) | 9 (10%) | 2 (2%) | - |
| Fatigue | 15 (17%) | - | - | - |
| Breast edema | 7 (8%) | - | - | - |
| Breast pain | 4 (4%) | - | - | - |

Table 1 - Acute Toxicity Observed from Study NYU 03-30

Longer follow up is required to assess local control, late toxicity, and to determine cosmetic results. Because of blood collection, once sufficient time has elapsed to measure late effects, the study will enable us to explore associations between specific genomic profiles and the

occurrence of fibrosis (Formenti 2005). In addition, this trial generated preliminary data on dose sparing to the heart and lung when patients are treated prone (Darby, McGale et al. 2005).

# 2.3 Rationale for Prone Radiotherapy: NYU 05-181

Despite the demonstrated feasibility and advantages of the prone set up, in our experience of more than 3,000 cases, occasional patients appear to be better treated supine, in order to optimally spare the heart and lung. Since no obvious clinical characteristics predict for this exception, NYU led a subsequent prospective effort of comparing supine versus prone breast setup in a consecutive cohort of 200 right and 200 left breast cancer patients. Again, intensity modulated radiotherapy with an accelerated, daily concomitant boost approach was used, the same regimen originally pilot-tested for prone IMRT. NYU Protocol 05-181, "Accelerated Intensity Modulated Radiation Therapy (AIMRT) to the Breast after Segmental Mastectomy: Identification of Optimal Individual Positioning" was opened in 2005 to pre- and postmenopausal women with stage 0 - IIB breast cancer who had received breast conserving surgery. Patient eligibility criteria included the requirement of at least 1 mm of margin, no more than 3 positive lymph nodes for breast cancer, at least two weeks post chemotherapy (if indicated), no history of prior or concurrent malignancy (within 3 years), and no history of active connective tissue disorders. Patients underwent CT simulation in both the prone and supine positions. Treatment followed in the optimal position that ensured the smallest volume of heart and lung respectively, in the target field.

From 2006 to 2009 the study met the planned accrual of 400 patients: 200 with left and 200 with right breast cancer. Results are summarized in Table 2. Among right breast cancer patients, the prone position was optimal in sparing lung volume in 98% (195/200), reducing the volume of lung in the treatment field by a mean 107 cc (SD 75, range 463,0). In the five patients treated supine, the choice for supine treatment was based on patient's preference since there was no significant difference in lung sparing between the two positions. For <u>left breast cancer</u> patients, the prone position was optimal in 85% (170/200), with lung volume reduced by a mean of 93 cc (SD 72, range 334, 9) and heart volume reduced by a mean of 11 cc (SD 23, range 0,220). However, in 15% of left breast patients, the best position was supine reducing the amount of heart in the treatment field by a mean of 6 cc (SD 8, range 0,41).

**Table 2 - Protocol 05-181 - Interim Results: Left/Right Breast Cancer by Supine/Prone Positioning** 

| | Supine | Prone | Total |
|-------|--------|-------|-------|
| Left | 30 | 170 | 200 |
| Right | 5 | 195 | 200 |

The experience gathered from the NYU 05-181 study provides support for all patients to first undergo a CT simulation in the prone position when the breast is to be irradiated. An additional supine set up will be attempted only if the dosimetry information derived from prone planning

Protocol Type / Version # / Version Date Version 5.4 06/30/2017

reveals that it exceeds the following normal tissue dose constraints:

- a. Heart:  $\geq$  5% of the heart volume receives greater than 5 Gy.
- b. Ipsilateral lung:  $\geq 15\%$  of the ipsilateral lung receives greater than 10 Gy.
- c. Contralateral lung: >15% of the contralateral lung receives greater than 5 Gy.

# 2.4 Rationale for Treating Axillary Level III and Supraclavicular Nodes

After breast surgery and an adequate axillary dissection (i.e., at least 8 nodes retrieved in the axillary dissection specimen from level I and II) it is possible to identify patients with 1 - 5 positive nodes who require radiotherapy to both the indexed breast/chest wall and the draining nodal stations that the surgeon did not include in the traditional level I - II axillary dissection, i.e., level III and supraclavicular stations. We are proposing to test a new technique that extends prone set up to also include these lymph node regions.

Limiting treatment to the supraclavicular fossa and level III axilla in patients with an adequately dissected axilla is supported by several published studies. Regional nodal recurrences are rare (occurring in 1 - 5%) in patients with early stage invasive breast cancer who have undergone breast conserving therapy (Fisher, Anderson et al. 2002; Moran and Haffty 2002; Harris, Hwang et al. 2003). Several institutions choose to treat only the level III axilla and supraclavicular nodal stations in patients who have undergone surgical treatment of level I/II axilla. This technique was documented recently by Liengsawangwong, who utilized CT-delineated nodal stations to improve target coverage of SCV and level III axillary nodes (Liengsawangwong, Yu et al. 2007) in patients who had undergone axillary level I/II dissection and were found to have positive lymph nodes.

Locoregional recurrences have been extensively studied in post-mastectomy patients as well. After chest wall recurrences, nodal failures in the undissected axillary level III or supraclavicular fossa are the second most common type of regional recurrence and occur more commonly in patients with four or more positive lymph nodes (Table 3) (Taghian, Jeong et al. 2004).

Table 3 - Locoregional Recurrence Rates in Post-mastectomy Patients without Radiotherapy

| Number LN+ | 1-3 LN+ (%) | ≥ 4 LN+ (%) | Median No. of LN Dissected | Chemotherapy Used |
|---|---|---|---|---|
| Danish trial 82b <sup>6</sup> | 30 | 42 | 7 | CMF |
| Danish trial 82c <sup>7</sup> | 31 | 46 | 7 | CMF |
| Canadian <sup>5</sup> | 33 | 46 | 11 | CMF |
| ECOG9† | 13 | 29 | 15 | CMF |
| MDA <sup>10</sup> ‡ | 14 | 25-34 | 17 | Doxorubicin based |
| IBCSG,11† premenopausal | 19.7§ | 30-38\$ | ≈15¶ | CMF** |
| IBCSG,11† postmenopausal | 16§ | 29-35\$ | ≈15¶ | CMF or tamoxifentt |
| NSABPt | 13 | 24-32 | 16 | Doxorubicin/CMF‡‡ |

Abbreviations: LN, lymph nodes; LN+, positive lymph nodes; CMF, cyclophosphamide, methotrexate, and fluorouracil; ECOG, Eastern Cooperative Oncology Group; MDA, M.D. Anderson Cancer Center; IBCSG, International Breast Cancer Study Group; NSABP, National Surgical Adjuvant Breast and Bowel Project.

The impact of extracapsular extension on outcome of post-mastectomy patients is controversial. Some studies report higher risk of distant recurrence, but no change in locoregional recurrence (Donegan, Stine et al. 1993) while others document higher rates of locoregional recurrence in patients with extracapsular extension (Garg, Strom et al. 2004; Huang, Tucker et al. 2005).

There may be a subset of high-risk patients who would benefit from adjuvant radiotherapy to the entire previously-dissected axilla. For example, an axillary boost to treat levels I/II decreased nodal recurrence, although it did not affect overall survival in a cohort of breast cancer patients with ten or more positive lymph nodes treated with breast conservation therapy (Chang, Feigenberg et al. 2007).

In summary, for some patients, the toxicity of any nodal radiotherapy will outweigh the benefit, while other patients have superior outcomes when the entire axilla and supraclavicular fossa are treated. There is likely a subset of breast cancer patients who could benefit from the advantage of limiting nodal radiotherapy to axillary level III and supraclavicular nodes after adequate axillary level I/II lymph node dissection, without impairing their chances of loco-regional control. Based on the previously referenced studies, we propose utilizing an approach of limited nodal treatment in patients with invasive breast cancer treated by breast conservation therapy or mastectomy with one to five involved lymph nodes after adequate dissection of level I/II axilla. These patients could also be studied to explore the feasibility and safety of an accelerated regimen of 3 weeks to the prone breast (or chest wall), and level III and supraclavicular nodes.

#### 2.5 Late Radiation Effects and Assessment of Risk

For patients who require regional nodal irradiation, an accelerated regimen of three weeks is very appealing, but in the past it has generally been discouraged because of concerns regarding the morbidity of larger doses to normal tissue, including lymphedema and brachial plexus

Protocol Type / Version # / Version Date Version 5.4 06/30/2017

<sup>\*</sup>Fifteen-year actuarial rate.

<sup>†</sup>Ten-year cumulative incidence.

<sup>‡</sup>Ten-year actuarial rate.

<sup>§</sup>Rate of LRF ± DF calculated from Table 5 from Wallgren et al.11

<sup>||</sup>Rate of LRF ± DF for patients with four to nine LN+ and ≥ 10 LN+, respectively.

<sup>¶</sup>Forty-seven percent of patients had 15 or more lymph nodes removed.

<sup>\*\*</sup>All patients received at least three courses of CMF chemotherapy.

<sup>††</sup>All patients received at least three courses of CMF chemotherapy or tamoxifen for 1 to 5 years.

<sup>‡‡</sup>The percentage of patients who received doxorubicin-based chemotherapy was 90.3%.

injury. The current protocol is likely to overcome some concerns of lymphedema by avoiding irradiation of the axillary stations where a surgical dissection was performed. Nevertheless, a field that includes axillary level III and the supraclavicular nodes will also include most of the ipsilateral brachial plexus, warranting cautious radiobiological modeling of late effects of radiotherapy to this target.

The severity of late effects is known to be dependent on both total dose and fraction size. In the linear-quadratic model, sensitivity to fraction size is expressed by the alpha/beta ratio, with a lower ratio indicating increased sensitivity. In a recent review, Kurtz summarized known alpha/beta values for tissues irradiated in breast cancer treatment (Table 4) (Kurtz 2005).

| Table 4 - A Review of Results Summarized by Kurtz et al. | | |
|---|---|---|
| End-point | Author (reference) | Alpha/beta (Gy) |
| Telangiectasia | Turesson et al. [14] | 4.2 |
| Chest wall fibrosis | Bentzen et al. [6] | 1.9 |
| Shoulder stiffness | Bentzen et al. [5] | 3.5 |
| Brachial plexus injury | Powell et al. [12] | 1.5-2.0 |
| Rib fractures | Overgaard [11] | 1.8-2.8 |
| Breast cosmesis<br>(fibrosis) | Van Limbergen<br>et al. [16] | 2.5 |

Due to low alpha/beta ratios for most of these tissues, it is possible that higher rates of late complications could be observed with an accelerated regimen. To clinically evaluate the impact of hypofractionation on brachial plexus injury, Powell et al. reported their experience with an accelerated schedule in a seminal paper published in 1990, describing the late effects of a group of 449 patients irradiated to the breast and regional lymph nodes with mean brachial plexus dose 45.9 Gy in 15 fractions (3 Gy per fraction) versus 54 Gy in 30 fractions (1.8 Gy per fraction) (Powell, Cooke et al. 1990). He noted a cumulative actuarial incidence of radiation-induced brachial plexus injury at 5.5 years of 5.9% versus 1.0% for the large and small fraction size group, respectively. It is important to note that the dose was higher than our proposed dose of 40.50 Gy given in 2.7 Gy daily fractions and that the fields included the entire axilla.

Lymphedema is another late complication sensitive to fraction size. Hayes documented rates of lymphedema in 2,579 patients followed at a single institution who underwent breast conservation therapy between 1970 and 2005. In patients receiving radiotherapy to the breast, breast + SCV, and breast + SCV + axillary boost, lymphedema occurred in 16%, 23%, and 31%, respectively (Hayes, Freedman et al. 2008). In a large phase III randomized trial, 46% of mastectomy patients experienced arm swelling at some point after radiotherapy (Deutsch, Land et al. 2008). For radical mastectomy patients, total mastectomy and radiotherapy patients, and total mastectomy patients in this trial, arm edema was recorded at least once in 58.1%, 38.2%, and 39.1% of patients, respectively (p < 0.001) and at last recorded measurement in 30.7%, 14.8%, and 15.5%, respectively (p  $\leq$  0.001). We anticipate that reduction of the size of the field for nodal radiation will reduce rates of lymphedema despite an accelerated treatment regimen.

Most patients experience lymphedema within the first years after treatment, but it can continue to increase in severity for more than five years after treatment in over 50% of patients (Bar Ad, Cheville et al. 2009). Therefore, subjects will need to be carefully followed for progressive lymphedema, for at least five years after radiotherapy is completed.

# 2.6 Dose Selection for Treating Breast and Nodal Stations

The linear-quadratic model (Lea 1942) can be used to determine whether the proposed IMRT protocol should result in a roughly equal probability of tumor control compared with a standard schedule, but without increasing the potential for normal tissue damage. The equation describing the single dose survival curve (Douglas and Fowler 1976) using this model is

$$-\ln S = (\alpha D + \beta D^2)$$

where S is the surviving fraction, D is the total dose and  $\alpha$  and  $\beta$  are tissue specific parameters. If the total radiation dose is delivered in a series of n fractions of dose d, rather than a single exposure, then the surviving fraction can be described as

$$-\ln S = n(\alpha d + \beta d^2)$$

which can be called the biological effect E. This equation can be rewritten as

$$E = (nd)(\alpha + \beta d) = (\alpha)(nd)(1 + d/\alpha/\beta)$$

If this equation is divided through by  $\alpha$ , then  $E/\alpha = (nd)(1+d/\alpha/\beta)$ . The quantity  $E/\alpha$  has been termed the biologically effective dose (15) or BED that is similar to the previously suggested extrapolated response dose (Barendsen 1982).

Hence,

BED = 
$$(nd)(1+d/\alpha/\beta)$$

This equation was used to calculate the BEDs for early and late responses, and tumor control for a standard schedule representing twenty-three 2 Gy fractions delivered once per day to the whole breast plus seven 2 Gy boost fractions to the tumor bed over a 39 day period. The proposed AIMRT schedule consists of fifteen IMRT fractions of 2.7 Gy to the whole breast and regional nodes and 3.2 Gy to the tumor bed delivered over an 18-day period. These calculations assume full repair takes place during the 24-hour or greater interval between fractions. Table 5 lists the BEDs for tumor control in addition to the early responses, erythema and desquamation, as well as the late responses, telangiectasia and fibrosis. The  $\alpha/\beta$  values used for these computations were reported in previous studies (Steel, Deacon et al. 1987; Matthews, Meeker et al. 1989; Turesson and Thames 1989; Thames, Bentzen et al. 1990; Archambeau, Pezner et al. 1995; Yamada, Ackerman et al. 1999).

**Table 5 - Biologically Effective Doses** 

| Normal Tissue Responses | | | | |
|---|---|---|---|---|
| | $\alpha/\beta$ | Standard | Standard | AIMRT |
| | (Gy) | Schedule | Schedule | Schedule |
| | | (2 Gy x 23 | (2 Gy x 25 | (2.7 Gy x 15 |
| | | in 39 days) | in 39 days) | in 18 days) |
| Brachial plexus injury | 2 | 92 Gy <sub>2</sub> | 100 Gy <sub>2</sub> | 95 Gy <sub>2</sub> |
| Fibrosis | 2 | 92 Gy <sub>2</sub> | 100 Gy <sub>2</sub> | 95 Gy <sub>2</sub> |
| Telangiectasia | 4 | 69 Gy4 | 75 Gy4 | 68 Gy4 |
| Erythema | 8 | 58 Gy <sub>8</sub> | 63 Gy8 | 54 Gy <sub>8</sub> |
| Desquamation | 11 | 54 Gy11 | 59 Gy11 | 50 Gy11 |
| Tumor Control | | | | |
| | α/β | Standard | AIMRT | AIMRT |
| | (Gy) | Schedule | Schedule | Schedule |
| | | (2 Gy x 30 | (3.2 Gy x 15 | (2.7 Gy x 15 |
| | | in 44 days) | in 18 days) | in 18 days) |
| Tumor | 2 | 120 Gy <sub>2</sub> | 125 Gy <sub>2</sub> | 95 Gy <sub>2</sub> |
| Tumor* | 2 | 116 Gy <sub>2</sub> | 125 Gy <sub>2</sub> | 95 Gy <sub>2</sub> |
| Tumor | 4 | 90 Gy4 | 86 Gy4 | 68 Gy4 |
| Tumor* | 4 | 86 Gy <sub>4</sub> | 86 Gy <sub>4</sub> | 68 Gy <sub>4</sub> |
| Tumor | 10 | 72 Gy <sub>10</sub> | 63 Gy <sub>10</sub> | 51 Gy <sub>10</sub> |
| Tumor* | 10 | 68 Gy <sub>10</sub> | 63 Gy <sub>10</sub> | 51 Gy <sub>10</sub> |

<sup>\*</sup>Taking into account cell proliferation during the course of treatment.

In terms of normal tissue responses, it can be observed from Table 5 that the BED values for the IMRT treatment are generally lower than the BEDs for the standard treatment for the early responses of erythema and desquamation. In addition, the BEDs are similar for the late responses of telangiectasia and fibrosis and brachial plexus injury. Hence, it would appear unlikely that the IMRT treatment will result in a greater risk of complications compared with the standard protocol.

With respect to tumor control, the classic dilemma typically encountered when a hypofractionated protocol is substituted for a standard treatment plan, is either a reduced probability of tumor control or an increased risk for late complications. This is due to the observation that fractionation generally results in greater sparing of late responding tissues compared with tumors. This finding is reflected in the relatively large  $\alpha/\beta$  values derived for tumors and small  $\alpha/\beta$  values for late responses (Thames and Hendry 1987).

In contrast to this generalization, evidence exists that breast cancer cells display a relatively low  $\alpha/\beta$ . This comes from in vitro studies in which  $\alpha/\beta$  values determined for breast cancer cell lines were generally about 4 Gy (Steel, Deacon et al. 1987; Matthews, Meeker et al. 1989; Yamada, Ackerman et al. 1999). The way in which this problem is diminished for this study is **Protocol Type / Version # / Version Date** Version 5.4 06/30/2017

through the use IMRT to limit the dose to the whole breast. Therefore, for the AIMRT protocol, the tumor bed will receive 3.2 Gy per fraction, whereas the breast and level III and supraclavicular will receive 2.7 Gy per fraction.

An even lower  $\alpha/\beta$  of 2 Gy can be calculated using the results of a prospective randomized trial (Baillet, Housset et al. 1990) in which a standard treatment of twenty-five 1.8 Gy fractions resulted in approximately the same level of tumor recurrence as a hypo-fractionated protocol of two 4.5 Gy plus two 6.5 Gy fractions. Therefore, if it is assumed that the BEDs for the two treatments were roughly equal, this yields an  $\alpha/\beta$  value of 2 Gy. Although there is evidence in the papers cited to support the use of these relatively low  $\alpha/\beta$  values for BED calculations, tumors on average exhibit greater  $\alpha/\beta$  values in the range of 10 Gy (Williams, Denekamp et al. 1985; Thames and Hendry 1987).

Viewing the results of the BED calculations for tumor control presented in Table 5, if the  $\alpha/\beta$  values are assumed to be in the range of 4 - 10 Gy, then there would appear to be only a small loss in BED for the AIMRT treatment, while for the 2 Gy  $\alpha/\beta$  value, the BED value for the alternate treatment actually is greater than the standard. In addition, it should be noted that the hypo-fractionated treatment also represents an accelerated protocol in which the total dose is delivered in only 18 days. Therefore, little or no tumor proliferation is likely to occur during the course of this proposed treatment as opposed to the standard treatment in which it is probable that tumor proliferation will take place thereby decreasing the chances for tumor control.

In order to take into account tumor proliferation for the BED calculation, it can be estimated that the number of clonogenic cells in the tumor (N) is related to the initial number of clonogens  $(N_0)$  by the expression

$$ln(N/N_0) = \lambda(T-T_k)$$

where  $\lambda$  is a constant related to the potential doubling time  $T_{pot}$  of the tumor by the expression,  $\lambda = \ln 2/T_{pot}$ , T is the total treatment time, and  $T_k$  (the "kick-off" time) is the time at which accelerated repopulation begins (15,26) (Travis and Tucker 1987; Fowler 1989). Note, this relationship is only valid for values of T greater than  $T_k$ . Therefore,

$$ln(N/N_0) = (ln2/T_{pot})(T-T_k)$$

Hence, the biological effect for a fractionated treatment should be *decreased* to take into account the increase in the number of cells due to repopulation and becomes:

$$E = n (\alpha d + \beta d^2) - (\ln 2/T_{pot})(T - T_k)$$

If this equation is divided through by  $\alpha$ , then the BED equation results and is given by

$$E/\alpha = [(nd) (1 + d/\alpha/\beta)] - [ln2(T-T_k)/\alpha(T_{pot})]$$

Hence, it is necessary to determine values for  $\alpha$ , the initial slope of the cell survival curve, as well as for  $T_{pot}$  and  $T_k$ . However, this may be either difficult or impossible to accomplish. Therefore, estimates are often made for these values in order to calculate the BED. For the purpose of these calculations, values of 0.3 for  $\alpha$ , (Steel, Deacon et al. 1987; Matthews, Meeker et al. 1989) 13 days for  $T_{pot}$  (Stanton, Cooke et al. 1996; Haustermans, Fowler et al. 1998) and 21 days for  $T_k$  were used. However, it must be stressed that the actual values for any given patient may differ significantly. Nevertheless, an effort was made to correct for tumor proliferation even though these calculations may be somewhat imprecise, as they still provide a better estimate of BED than a determination of this parameter performed in the absence of any cell proliferation correction factor.

As presented in Table 5, the equation above which incorporates a cell proliferation correction factor produces small decreases in the BEDs for the standard treatment. Therefore, taking into consideration tumor proliferation during treatment, the IMRT schedule results in BED values greater to or equal to the standard treatment for  $\alpha/\beta$  values of either 2 or 4 Gy and is only slightly lower when a 10 Gy  $\alpha/\beta$  value is used. In addition, it must be kept in mind that there is a range of  $T_{pot}$  values for a population of tumors. Therefore, the accelerated nature of the AIMRT treatment may have a particularly beneficial effect for those patients whose tumors are characterized by relatively short  $T_{pot}$  values.

Of course, if cell proliferation is taken into account, this also diminishes the BEDs and lessens the severity of the anticipated early responses for the standard schedule compared with the AIMRT schedule. This should not affect late responses because the  $T_k$  is generally greater than the total treatment time for late responding tissues as compensatory proliferation usually does not begin until after completion of a standard protocol. However, even if the BEDs were decreased to take into account cell proliferation, this would probably result in only slightly diminished BEDs for erythema and desquamation for the standard schedule, resulting in BEDs comparable to the AIMRT schedule.

# 2.6.1 Rationale for this Approach

The proposed treatment approach entails radiotherapy to axillary level III and SCV, defined by CT imaging obtained in a prone position using IMRT technique. We anticipate that this will improve target coverage, toxicity, and tolerability for several reasons. First, by avoiding radiotherapy to level I and II axillary lymph nodes in a previously dissected axilla, we anticipate reduced risk of lymphedema. Additionally, treatment in the prone position has been shown to reduce dose to heart and lungs (Formenti, Gidea-Addeo et al. 2007), which may decrease late toxicity to these organs. Finally, while standard 3-field and 4-field techniques provide inadequate lymph node coverage in the prone position (refer to preliminary data in Section 2.6.2), use of IMRT technique will enable prone target coverage while maintaining low doses to normal tissues.

# 2.6.2 Preliminary Data

To evaluate the dosimetric feasibility of the prone IMRT treatment approach and to compare its dosimetric performance compared to other standard techniques, we explored six treatment planning techniques to target the breast and axillary level III and supraclavicular nodes.

The CT images of 10 breast cancer patients (7 left, 3 right) who underwent simulation in both prone and supine positions were used for planning. Supraclavicular and level III axillary lymph node regions, breast tissue, tumor bed, heart, and ipsilateral lung were manually contoured. Six treatment plans were created for each patient; all utilized tangential fields to target breast tissue. A three-dimensional conformal radiotherapy (3DCRT) plan with a single anterior-oblique field, a 3DCRT plan with anterior-oblique and posterior axillary boost fields, and an intensity-modulated radiotherapy (IMRT) plan were utilized to target regional nodes in both prone and supine positions. Dose-volume histograms were compared to evaluate lymph node coverage and normal tissue dose. Two-tailed student t-test was used to identify statistically significant differences between planning techniques. Nodal target and normal tissue doses from the six techniques are summarized below in Tables 6 - 8.

**Table 6 - Prone Compared to Supine Positioning** 

| | mean (st dev, range) | mean (st dev, range) | p-value |
|---|---|---|---|
| | 3-field supine | 3-field prone | |
| PTV-V50 | 53.96% (18.20, 25.70-75.00) | 34.10% (21.91, 4.50-73.10) | 0.0407559 |
| Lung-V40 | 14.70% (4.84, 8.30-24.40) | 3.81% (4.41, 0.10-14.40) | 0.0000530 |
| Lung-V20 | 22.98% (5.23, 16.50-33.80) | 9.52% (5.98, 2.10-21.20) | 0.0000434 |
| Lung-V5 | 31.57% (5.82, 24.00-42.10) | 13.57% (6.83, 4.90-27.90) | 0.0000056 |
| Heart-V20 | 0.15% (0.30, 0.00-0.80) | 0.04% (0.08, 0.00-0.20) | 0.2687512 |
| Heart-V5 | 0.72% (1.07, 0.00-2.70) | 0.38% (0.44, 0.00-1.20) | 0.3436903 |
| Spinal cord- | | | |
| Dmax | 1131.90 cGy (333.38, 782.00-1712.00) | 889.60 cGy (273.04, 263.00-1258.00) | 0.0922816 |
| | IMRT supine | IMRT prone | |
| PTV-V50 | 94.59% (0.32, 94.00-95.00) | 95.48% (0.69, 94.80-97.00) | 0.0016879 |
| Lung-V40 | 15.28% (3.06, 11.90-21.80) | 6.54% (1.98, 3.50-9.00) | 0.000005 |
| Lung-V20 | 27.22% (6.88, 18.60-37.80) | 12.48% (3.29, 8.20-17.90) | 0.0000089 |
| Lung-V5 | 43.73% (7.47, 32.30-56.90) | 24.18% ( 5.09, 19.50-33.40) | 0.0000021 |
| Heart-V20 | 0.12% (0.26, 0.00-0.70) | 0.37 (0.72, 0.00-2.00) | 0.3011538 |
| Heart-V5 | 0.62% (0.93, 0.00-2.40) | 0.93% (1.08, 0.00-3.70) | 0.6524424 |
| Spinal cord- | | | |
| Dmax | 3490.70 cGy (765.64, 1963.00-4266.00) | 2805.20 cGy (953.84, 1762.00-4112.00) | 0.0932683 |
| | 4-field supine | 4-field prone | |
| PTV-V50 | 60.77% (12.56, 36.90-83.50) | 38.93% (20.65, 1.80-78.60) | 0.0104802 |
| Lung-V40 | 12.29% (7.38, 0.70-25.30) | 5.59% (4.70, 0.00-15.60) | 0.0262689 |
| Lung-V20 | 20.53% (8.34, 2.20-34.10) | 10.93% (6.65, 2.10-26.30) | 0.0107219 |
| Lung-V5 | 29.78% (10.27, 5.60-43.70) | 16.40% (8.19, 5.90-36.50) | 0.0047406 |
| Heart-V20 | 0.50% (1.05, 0.00-2.80) | 0.06% (0.10, 0.00-0.20) | 0.2870816 |
| Heart-V5 | 1.84% (3.09, 0.10-8.50) | 0.53% (0.42, 0.20-1.20) | 0.2864321 |
| Spinal cord- | | | |
| Dmax | 836.20 cGy (225.60, 560.00-1258.00) | 739.10 cGy (134.95, 418.00-872.00) | 0.2580200 |

These results indicate that all 3DCRT plans had inadequate lymph node coverage, with mean planning target volume (PTV) V50 Gy 54% supine and 34% prone (3-field 3DCRT), and 61% supine and 39% prone (4-field 3DCRT). Compared to these techniques, IMRT significantly improved nodal coverage, with mean PTV V50 Gy 95% supine and 95% prone (p < 0.001, two-Protocol Type / Version # / Version Date Version 5.4 06/30/2017

tailed t-test). Prone positioning resulted in significantly lower ipsilateral lung doses: mean V20 Gy was 10% prone versus 23% supine (3-field 3DCRT, p < 0.001, two-

tailed t-test); 21% supine versus 11% prone (4-field 3DCRT, p = 0.01, two-tailed t-test); and 12% prone versus 27% supine (IMRT, p < 0.001, two-tailed t-test). Among the 7 left breast

Table 7 - Supine IMRT Compared to Supine 3F/4F

| Table 8 - Prone livik i | Compared to Prone 3F/4F | |
|-------------------------|-------------------------|---|
| | | • |

| | mean | mean | p-value | | Mean | mean | p-value |
|---|---|---|---|---|---|---|---|
| | 3-field supine | IMRT supine | | | 3-field prone | IMRT prone | |
| PTV-V50 | 53.96 | 94.59 | 0.0000014 | PTV-V50 | 34.10 | 95.48 | 0.000001 |
| Lung-V40 | 14.70 | 15.28 | 0.7525528 | Lung-V40 | 3.81 | 6.54 | 0.0909352 |
| Lung-V20 | 22.98 | 27.22 | 0.1382071 | Lung-V20 | 9.52 | 12.48 | 0.1876868 |
| Lung-V5 | 31.57 | 43.73 | 0.0007318 | Lung-V5 | 13.57 | 24.18 | 0.0009626 |
| Heart-V20 | 0.15 | 0.12 | 0.8059355 | Hrt-V20 | 0.04 | 0.37 | 0.1577367 |
| Heart-V5 | 0.72 | 0.62 | 0.8108750 | Hrt-V5 | 0.38 | 0.93 | 0.2202274 |
| Spinal cord-Dmax | 1131.90 | 3490.7 | 0.00000005 | Cord-Dmax | 889.60 | 2805.20 | 0.0000091 |
| | 4-field supine | IMRT supine | | | 4-field prone | IMRT prone | |
| PTV-V50 | 60.77 | 94.59 | 0.000001 | PTV-V50 | 38.93 | 95.48 | 0.000001 |
| Lung-V40 | 12.29 | 15.28 | 0.2521097 | Lung-V40 | 5.59 | 6.54 | 0.5635124 |
| Lung-V20 | 20.53 | 27.22 | 0.0027134 | Lung-V20 | 10.93 | 12.48 | 0.5172072 |
| Lung-V5 | 29.78 | 43.73 | 0.0027134 | Lung-V5 | 16.4 | 24.18 | 0.0200405 |
| Heart-V20 | 0.5 | 0.12 | 0.4401863 | Hrt-V20 | 0.06 | 0.37 | 0.2744447 |
| Heart-V5 | 1.84 | 0.62 | 0.4509997 | Hrt-V5 | 0.53 | 0.93 | 0.2089303 |
| Spinal cord-Dmax | 836.2 | 3490.7 | 0.000000004 | Cord-Dmax | 739.1 | 2805.20 | 0.0000024 |

cancer patients, there was no statistically

significant difference in mean heart V20 Gy or V5 Gy (p > 0.05, two-tailed t test).

#### 2.7 Quality of Life Assessment

Quality of life (QOL) assessments will be performed by patients at regular intervals (i.e., baseline, last week of treatment, 45 - 60 days from starting radiotherapy and 2-year follow-up). Patients status post mastectomy will be asked to answer applicable questions only in the QOL assessment. This trial will use the QLB and QLF questionnaires from the RTOG.

The QLB and QLF questionnaires are derived from a validated integration of parts of the BCTOS and MOS SF 36. BCTOS is a validated questionnaire that measures cosmetic results based on patient self-reports. This brief self-report instrument has high reliability and validity, and has been used in a variety of previous studies on recovery from breast cancer treatment (Stanton, Krishnan et al. 2001). MOS SF36 is a common QOL questionnaire used in cancer patients (Shelbourne 1992; Ware and Sherbourne 1992).

#### 2.8 Measuring the Late Toxicities of Breast and Nodal Radiation

Hoeller et al. recently reported a careful comparison of The Radiation Therapy Oncology Group (RTOG) and Late Effects Normal Tissue Task Force subjective, objective, management, and analytic (LENT/SOMA) scores for late breast toxicity after radiation in a group of breast cancer patients (Hoeller, Tribius et al. 2003). In comparison, when LENT/SOMA criteria were used, telangiectasia and pigmentation were upgraded in 34% and 36% of patients, respectively, and

telangiectasia was downgraded in 45% of patients. Inter-observer variability was similar for both classification systems and ranged from Cohen's kappa 0.3 (retraction) to 0.91 (telangiectasia). The authors concluded that LENT/SOMA criteria seem to be the better tool in grading and recording late radiation toxicity as compared to the RTOG scale. Specifically, fibrosis scores correlated well with the LENT/SOMA scoring system (Spearman's rho 0.78, p = 0.01). The LENT/SOMA scoring system will be used in the reporting of late radiation morbidity in this protocol.

# 2.8.1 Quantitative Measurement of Thyroid Function

Patients undergoing radiotherapy for invasive breast cancer are at higher risk of hypothyroidism. One recent study documented hypothyroidism in 18% of patients with stage II/III invasive breast cancer who had undergone radiotherapy, compared to only 6% (p < 0.001) of an age-matched control group from the general population (Reinertsen, Cvancarova et al. 2009).

As such, patients will undergo thyroid function testing, including measurement of serum thyroid stimulating hormone (TSH) and free T<sub>4</sub> levels, at baseline and at yearly intervals after completion of radiotherapy.

# 2.8.2 Quantitative Measurement of Lymphedema

Patients will be assessed for lymphedema at baseline, end of treatment, and at yearly intervals after completion of radiotherapy. Arm circumference at sites 10 cm above and below the antecubital fossa will be obtained. Mild, moderate, and severe lymphedema is defined as a difference of 0.5 to 2 cm, 2.1 to 3 cm, and greater than 3 cm, respectively, of arm circumference at one or more measurement sites on the treated versus untreated side. Lymphedema progression is defined as transition from lower to higher grade at any time point. Similar lymphedema classification systems have been used in previously published studies (Keramopoulos, Tsionou et al. 1993; Bar Ad, Cheville et al. 2009).

#### 2.8.4 Genetics of Radiation-induced breast fibrosis

Since the most likely long-term toxicity of accelerated radiation is soft tissue fibrosis and skin telangiectasia the preliminary recognition of genetic predispositions to these complications enables the exclusion of high-risk carriers from the trials of accelerated/hypo-fractionated radiation. In other words, similar to the impact of pharmacogenomics in medical oncology, the field of radiation-genomics is also rapidly emerging, permitting identification of individuals with genetic predisposition to inferior repair of the damage caused by ionizing radiation.

A recent study from Quarmby et al. has shed some light on the genetic risk of developing breast fibrosis post-ionizing radiation. To investigate whether single nucleotide polymorphisms (SNP) of transforming growth factor beta-1 (TGF-beta1) were associated with the susceptibility of

breast cancer patients to severe radiation-induced normal tissue damage, Quarmby et al. performed Polymerase Chain Reaction-Restriction Fragment Length Polymorphism (PCR-RFLP) assays for TGF-beta1 gene polymorphisms on DNA obtained from 103 breast cancer patients who received radiotherapy (Quarmby, Fakhoury et al. 2003). The G-800A, C-509T, T+869C and G+915C polymorphic sites were examined, and genotype and allele frequencies of two subgroups of patients were calculated and compared. The investigators found that the less prevalent -509T and +869C alleles were significantly associated with a subgroup of patients who developed severe radiation-induced normal tissue fibrosis (n = 15) when compared with those who did not (n = 88) (odds ratio = 3.4, p = 0.0036, and 2.37, p = 0.035, respectively). Furthermore, patients with the -509TT or +869CC genotypes were between seven and 15 times more likely to develop severe fibrosis. These findings imply a role for the -509T and +869C alleles in the biological mechanisms underlying susceptibility to radiation-induced fibrosis.

#### 2.8.5 Blood Collection for Future Genomic Studies

The purpose of this portion of the study will be to collect blood from each subject accrued to the study for the  $-509C \rightarrow T$  and  $+869T \rightarrow C$  TGF- $\beta1$  polymorphisms that have been reported to be correlated with the development of fibrosis following radiotherapy for treatment of breast cancer (Quarmby, Fakhoury et al. 2003).

It is first important to note that Dr. Rosenstein's (co-investigator) laboratory has extensive experience in the detection of genetic alterations using Denaturing High Performance Liquid Chromatography (DHPLC) (Atencio, Iannuzzi et al. 2001; Iannuzzi, Atencio et al. 2002; Bernstein, Teraoka et al. 2003). In addition, our group is part of the WECARE consortium of four laboratories that is in the process of using DHPLC to screen 2100 breast cancer patients for mutations and SNPs in a variety of genes associated with DNA repair and radiation responses. Hence, our laboratory has substantial expertise performing genetic analysis using DHPLC and will therefore be able to immediately implement this portion of the project.

For the purpose of this trial blood will be collected to enable future genomic analysis for this polymorphism to explore association with the incidence of grade 3 and 4 late complications at 3 years follow up and for other related research studies. Methods details of DHPLC are covered in Section 10.4.

#### 3 PATIENT SELECTION

# For Cohort A: Include patients who have undergone SLNB without completion ALND)

- 3.1 Inclusion Criteria
  - 3.1.1 Pre- or post-menopausal women with stage II III breast cancer (AJCC 2002)
  - 3.1.2 Biopsy-proven invasive breast cancer, excised with negative margins of at

- least 1 mm
- 3.1.3 Status post segmental mastectomy or mastectomy and axillary node dissection with removal of at least 8 nodes
- 3.1.4 One to 5 involved lymph nodes identified at axillary staging
- 3.1.5 At least 2 weeks from last chemotherapy or before chemotherapy
- 3.1.6 No more than sixty days from final surgery to simulation if no systemic therapy (includes chemotherapy and Hormonal therapy) is given
- 3.1.7 Patient needs to be able to understand and demonstrate willingness to sign a written informed consent document

#### 3.2 Exclusion Criteria

- 3.2.1 Previous radiation therapy to the ipsilateral breast
- 3.2.2 More than 5 involved nodes identified at axillary staging
- 3.2.3 Current treatment for active connective tissue disorders, such as lupus or scleroderma
- 3.2.4 Pregnant or lactating women
- 3.2.5 Less than 35 years old
- 3.2.6 Prior concurrent malignant other than basal or squamous cell carcinoma or carcinoma in situ of cervix unless disease free > 3 years

#### 4 REGISTRATION PROCEDURES

#### 4.1 General Guidelines

Patients will have completed all breast surgical procedures prior to accrual into this protocol in order to establish eligibility criteria. Final pathology margins must be at least 1 mm in all directions to be eligible. The patient may undergo re-excision if the initial margins are involved or close (< 1 mm). If the patient meets the eligibility criteria after re-excision, she may be entered into the left or right breast cancer strata. AJCC staging criteria will be used to identify clinical stage II - III breast cancer patients' eligible to this study. All eligible women who are referred to the Radiation Oncology Department at NYU School of Medicine for radiation following surgery for breast cancer will be offered the opportunity to participate in this experimental protocol.

# 4.2 Registration Process

Before any protocol specific procedures can be carried out, investigators/staff will fully explain the details of the protocol, the study procedures and the aspects of patient privacy regarding research information. Patients or their legal guardians will be provided a comprehensive explanation of the proposed treatment including the type of therapy, the rationale for treatment on the protocol, alternative treatments that are available, any known adverse events, the investigational nature of the study and the potential risks and benefits of the treatment. The informed consent document will meet all requirements of the Institutional Review Board (IRB). All subjects/patients are informed in the consent that participation or refusal to participate in the

research study will not affect any of the clinical treatment or services to which they would otherwise be entitled.

The physicians who may obtain informed consent are listed on the title page of this protocol. The informed consent form will be signed by the participant and the registering physician. Once signed, a copy will be given to the patient and one will be maintained with the patient's medical record. Once eligibility is confirmed and informed consent is documented, the patient will be registered by the study coordinator/data manager.

#### 5 TREATMENT PLAN

# 5.1 General Concomitant Medication and Supportive Care Guidelines

During radiation treatment, all patients will be prescribed daily application of Calendula lotion or equivalent, to prevent skin dryness and reduce erythema.

# 5.2 Duration of Therapy

The treatment will consist of 15 fractions, with one fraction daily for five days a week, for 3 consecutive weeks.

# 5.3 Duration of Follow-up

Patients will be seen for follow-up at 45 - 60 days from first radiotherapy treatment, and then yearly for up to 5 years.

#### 5.4 Alternatives

At the time of study accrual, all patients will be offered access to standard six weeks radiotherapy, including 5 weeks of treatment to the whole breast or chest wall and regional lymph nodes using a standard 4-field plan, followed by a boost to the tumor bed or scar if required.

# 5.5 Compensation

No compensation is available for participating in the study.

#### 6 SURGERY

Patients will have completed all breast cancer surgical procedures prior to accrual into this protocol in order to establish eligibility criteria. Final pathology margins must be at least 1 mm in all directions to be eligible. The patient may undergo re-excision if the initial margins are involved or close (< 1 mm). If the patient meets the eligibility criteria after re-excision, she may be entered onto the study. Patients must also undergo lymph node dissection of axillary levels

Protocol Type / Version # / Version Date Version 5.4 06/30/2017

I/II with removal of at least 8 nodes.

#### 7 RADIOTHERAPY SPECIFICATIONS

# 7.1 Treatment Planning using Hybrid IMRT Technique

In the context of a Phase I/II prospective study, this protocol will test whole breast and regional nodal radiotherapy using a hybrid approach. Patients will receive whole breast radiotherapy in a prone position with a concomitant daily boost to the tumor bed over three weeks, a technique which has previously been evaluated in over 500 patients (NYU 03-30 and NYU 05-181) and has shown excellent tolerance and results. In addition, an intensity modulated radiation therapy (IMRT) technique will be used to deliver concomitant radiotherapy to axillary level III and supraclavicular lymph nodes. In patient Cohort A, axilliary levels I and II will also be part of the radiation target. Patients status post mastectomy will receive whole reconstructed breast/chest wall radiotherapy and nodal irradiation. A concomitant boost to the scar region will be offered only to patients without reconstruction.

# 7.2 Dose Specification

Patients will receive 15 daily radiation fractions of 2.7 Gy, Monday to Friday for three weeks, to the entire breast/chest wall and axillary level III and supraclavicular nodes with a daily concomitant boost of 0.5 Gy to the tumor bed, for a total daily dose of 3.2 Gy to the tumor bed (2.7 Gy + 0.5 Gy). The overall dose will be 40.5 Gy to the breast/chest wall, axillary level III and supraclavicular nodes, and 48.0 Gy to the tumor bed.

#### 7.3 CT Simulation

All patients will be CT scanned in the prone position on a specially designed board that allows the indexed breast tissue to fall freely below the board, granting unobstructed access to the breast through radiation ports from multiple beam angles. CT slice thickness should be 3.75 mm or less. Prior to the patient lying prone on the table for scanning, the borders of the breast/chest wall fields will be marked with radio-opaque CT fiducial markers. These markers will be used to outline the breast/chest wall treatment volume according to conventional treatment guidelines. Borders of the fields will be set medially at mid-sternum, laterally at the anterior edge of latissimus dorsi, superiorly at the bottom of the clavicular heads and inferiorly 2 cm from the infra-mammary fold. Patients will be tattooed with leveling marks for setup alignment with room lasers and for positioning the isocenter of the beams. A tattoo will be placed on the lateral breast tissue as a landmark for planning and positioning. Patients status post mastectomy will also be simulated prone with similar field borders. In addition, the chest wall scar will carefully be marked with radio-opaque CT fiducial markers.

Contouring of breast tumor bed, axillary level III nodes, supraclavicular nodes, indexed and contralateral breast tissue, ipsilateral brachial plexus, esophagus, heart, right and left lung, spinal cord, spinal cord plus 5 mm margin and right and left lobes of the thyroid will be

performed in order to guide beam arrangement and optimal normal tissue avoidance. In patients who have undergone pre-operative breast MRI, the breast glandular tissue will be contoured with the help of a radiologist co-investigator (Drs. Moy and Newburg), to better inform the design of the treatment fields.

The patient will be CT scanned and treated in the supine position if the patient cannot lie prone, or if the prone plan fails to satisfy the dose constraints specified in Section 7.5.6

# 7.4 Target Delineation

- 7.4.1 The physician designs tangent fields to encompass the whole breast. The PTVBreast is created from the 50% isodose line associated with the tangent fields. Technically this is accomplished by converting the 50% isodose level to a structure, smoothing and then removing parts extending outside the 50% isodose structure with an additional 0.6 cm margin. The PTVBreast volume overlapping the heart and lung is excluded.
- 7.4.2 PTVTumor is the tumor bed, as identified on CT with an additional 1.0 cm 3D margin. Post-mastectomy PTVTumor is the tumor bed and depending on clinical judgement may or may not include the scar.
- 7.4.3 PTVTumor Eval is the PTVTumor cropped 0.6 cm from the skin.
- 7.4.3 PTVNodes includes axillary level III and supraclavicular lymph nodal regions as identified on CT with an additional 0.5 cm 3D margin. For patients in Cohort A PTVNodes will include axillary levels I-III and supraclavicular nodal regions as identified on CT with an additional 0.5 cm 3D margin, However, the PTV will not be expanded medially to better spare the esophagus.
- 7.4.4 PTVNodesEval is the PTVNodes cropped 0.6 cm from the skin.

#### 7.5 Technical Factors

- 7.5.1 Dose calculations will include heterogeneity corrections.
- 7.5.2 Whole Breast fields 3D tangents plus IMRT tangents
  - 1. The prone position requires careful placement of the isocenter during planning to avoid collision between the gantry and the breast board, couch, or patient.
  - 2. 3D tangents deliver nominally 67% of the whole breast dose, using 6 MV photons and including 2-3 cm flash. The fields are wedged and weighted to obtain a uniform dose distribution, normalized to allow approximately 105% maximum dose. 16 MV photons may be used for patients with large separations to reduce magnitude of dose maximum.
  - 3. IMRT tangents deliver nominally 33% of the whole breast dose, using 6 MV photons and including 2-3 cm flash. The 3D tangents are used as a base for optimization.

# 7.5.3 Axillary level I-III and supraclavicular nodes (PTVNodes)

1. Three or more IMRT fields.

#### 7.5.4 PTVTumor fields

- 1. Non-coplanar beam arrangement is encouraged, but not required.
- 2. Integrated boost within the IMRT tangents is allowed.
- 3. Electron therapy may be utilized.
- 4. No photon beam will be directed toward heart, lung, contralateral breast, or thyroid
- 5. Inclusion of soft tissue not irradiated by the whole breast tangents is allowed to aid in target coverage.
- 6. If the PTVTumor, as visualized in the beams-eye-view (BEV), is within 1 cm of the body surface, 1 cm of flash will be added to the field(s), painting fluence for IMRT fields.

# 7.5.5 IMRT Optimization

IMRT optimization is performed either by using the 3D tangents plan as a base plan for all IMRT fields, or by using a plan with all tangent fields (IMRT and 3D) as a base for the IMRT nodal fields. Regardless, a single plan is created with 3D breast tangent fields, IMRT breast tangent fields, boost fields if used, and IMRT axillary level III and supraclavicular nodal fields.

#### 7.5.6 Dose Constraints

The dose constraints below represent acceptance criteria for the resulting dose distribution

- 1. Target volume dose constraints:
  - PTVTumor: V 48 Gy > 98%
  - PTVBreast: V  $40.5 \text{ Gy} \ge 95\%$
  - PTVNodesEval: V 38.5 Gy > 95%
- 2. Normal tissue dose constraints:
  - a. Heart: V 5 Gy < 5%
  - b. Ipsilateral lung: V 10 Gy < 20%
  - c. Contralateral lung: V 5 Gy < 15%
  - d. Spinal cord: 37.5 Gy maximum
  - e. Spinal cord plus 0.5 cm margin: 40 Gy maximum
  - f. Thyroid: contralateral lobe 15 Gy maximum
  - g. Esophagus: V 30 Gy < 50%, 40.5 Gy maximum
  - h. Ipsilateral brachial plexus: 42 Gy maximum
  - i. Contralateral breast: Efforts should be made to keep the contralateral breast completely outside the primary beams

# 7.6 Portal Imaging

Portal images of orthogonal setup fields will be acquired on days 1, 2, and 3 then weekly thereafter. In addition, portal images will be acquired of each treatment field (except where geometrically impractical) during the first three days of treatment.

Cone beam CT (CBCT) of the nodal region will be acquired once on a day when orthogonal setup fields are imaged. No alignment adjustment will be made based on the CBCT.

# 8 DOSE MODIFICATIONS AND STOPPING CRITERIA

#### 8.1 Dose Modification

In case of grade 3 acute skin toxicity occurring during the course of the 3-week treatment, the dose per fraction of the remaining treatment fractions will be reduced to 2 Gy/fraction until completion.

# 8.2 Stopping Criteria

Regional nodal recurrences occur in 1 - 5% of patients with early stage breast cancer who have undergone mastectomy or breast conserving therapy (Fisher, Anderson et al. 2002; Moran and Haffty 2002; Harris, Hwang et al. 2003). While most nodal recurrences occur within the first five years after treatment, nodal recurrences have been documented for more than twenty years after completion of treatment (Lukens, Vapiwala et al. 2009).

Based on this data, a stopping rule for regional node recurrences will be implemented with an evaluation after every 21 patients are observed for at least 1 year post treatment. The schema is described in Section 14. This rule allows early stopping based on an excess of incidence of regional node recurrences (greater than 5% of patients).

# 9 ADVERSE EVENTS: LIST AND REPORTING REQUIREMENTS

#### 9.1 Adverse Events and Potential Risks List

Expected toxicities include fatigue and skin reactions within the radiation field. Erythema, dry and moist desquamation of the skin will be recorded weekly. Breast edema and tenderness are additional possible acute side effects. Acute ( $\leq$  60 days after first day of treatment) and late toxicity (> 60 days after first day of treatment) will be reported as scheduled in the study calendar. This study will utilize the descriptions and grading scales as described in *Common Terminology Criteria for Adverse Events v3.0 (CTCAE)* for acute toxicity and in the LENT/SOMA classification for late toxicities (appendix 1). Toxicities will be tracked using the Toxicity Tracking Form (appendix 2).

# 9.2 Expedited Adverse Event Reporting

Expedited AE reporting will utilize the descriptions and grading scales as described in *Common Terminology Criteria for Adverse Events v 3.0 (CTCAE)*. SAEs that occur in this study must be promptly reported to the study P.I. (Dr. Carmen Perez) as well as to the NYU IRB and to the NYU Clinical Trials Office for reporting to the NYUCI Data Safety Monitoring Committee.

# 9.3 Routine Adverse Event Reporting Guidelines

The IRB Reportable Events Forms (available electronically at http://irb.med.nyu.edu/sites/default/files/irb2/app.reportable.event\_.2012.03.07.docx) will be used for all adverse events

#### 10 CORRELATIVE/SPECIAL STUDIES

# 10.1 Blood Collection for TGF-beta 1 Polymorphism Determination

Approximately 30 mL of blood will be obtained by venipuncture once before starting treatment and once on the last day of treatment, after the last dose of radiation. The specimen will be aliquoted and stored for future testing of other polymorphisms and other related research studies.

# 10.2 Lymphocyte Isolation, DNA Extraction, PCR Amplification and DNA Sequencing

The lymphocyte isolation and DNA extraction and DHPLC procedures will be performed as previously described (Iannuzzi, Atencio et al. 2002) using the Wave<sup>TM</sup> DNA Fragment Analysis System manufactured by Transgenomic. Any samples that appear, based upon the DHPLC screening, to be homozygous for either the –509C $\rightarrow$ T or +869T $\rightarrow$ C TGF-β1 polymorphism, will be subjected to DNA sequencing using an automated DNA sequencer.

#### 10.3 Test Method

The products of the PCRs will be subjected to DHPLC analysis with the 96 well plate placed in the DHPLC apparatus. The Wave<sup>TM</sup> DNA Fragment Analysis System (Transgenomic), which will be used for this project, represents a complete unit for the automated DHPLC analysis of PCR products using a DNASep cartridge specifically designed for separation of DNA fragments. DHPLC is a high throughput technique in which large numbers of DNA samples can be rapidly screened for base sequence alterations and relies upon the physical changes in DNA molecules induced by mismatched heteroduplex formation during reannealing of wild type and mutant DNA.

In this method, a portion of a gene is amplified using standard PCR conditions and the products analyzed using DHPLC. Material from a homozygous sample will only form one species, the wild-type homoduplex. However, when the PCR products produced from a sample **Protocol Type / Version # / Version Date** Version 5.4 06/30/2017

heterozygous for a base sequence alteration are heated to 95°C, and then slowly cooled, the DNA strands separate and randomly reanneal to form a mixture of four species; a mutant homoduplex, two heteroduplexes and a wild type homoduplex. When mutant and wild-type DNA strands reanneal to form a heteroduplex, the molecule is physically altered. At the region of base pair mismatches, a "bubble" forms yielding a short linear region of single-stranded DNA. This structural alteration provides the basis for separation of heteroduplex from homoduplex species and ultimately identifies samples with mutant alleles. The basis of this technique is that by heating the column during separation, it is possible to partially denature the sample and elute the homoduplexes and heteroduplexes separately. Heteroduplexes, having a greater percentage of single-stranded DNA than homoduplexes in the mismatch region at a given temperature, will elute first from the column. Therefore, if the DNA sample does not possess a base sequence alteration, only homoduplexes will form and there will be only one peak on the chromatogram representing the homogenous nature of the fragment. A sample that contains a heterozygous mutation will appear as 2, 3 or 4 peaks representing the two homoduplex and heteroduplex populations.

It is also important to note that samples homozygous for a polymorphic allele can readily be detected using DHPLC by adding a roughly equal amount of DNA to the PCR from a sample known to be homozygous for the normal allele, thus essentially creating a potentially "heterozygous" sample.

The first step in the process to detect the −509C→T and +869T→C TGF-β1 gene polymorphisms will be to design primers for amplification of these regions following which the DHPLC buffer and temperature conditions will be optimized for detection of these polymorphisms. For each sample, the PCRs will be performed first without the addition of DNA from a sample that is known to be homozygous for the normal allele, and then, depending upon the DHPLC results, with the addition of known wild type DNA.

For samples in which DNA homozygous for the normal allele was not added, one peak in the DHPLC will indicate it is homozygous for either the wild type or polymorphic allele, whereas multiple peaks will signify it is heterozygous. Next, the PCRs will be performed a second time for all of the putative homozygotes to determine for which allele they are homozygous. Thus, DNA homozygous for the normal allele will be added to the PCR. If there is still one peak in the DHPLC, this will indicate that it is homozygous for the normal allele, whereas if there are multiple peaks, this will signify that the subject is homozygous for the polymorphic allele. All samples which appear to be homozygous for the polymorphic allele will be subjected to DNA sequencing to confirm this assignment.

An important step in this process will be a determination of the appropriate amount of homozygous normal allele DNA to be added to the PCR. Therefore, a titration will be performed with different concentrations of DNA to determine the amount for clearest detection of a sample homozygous for the polymorphic allele.

# 10.4 Denaturing High Performance Liquid Chromatography (DHPLC)

The mutation screening technique to be used in this study will be denaturing high performance liquid chromatography or DHPLC (Huber, Oefner et al. 1993; Huber, Oefner et al. 1993; Kuklin, Munson et al. 1997; Oefner and Underhill 1998). DHPLC is a robust technique that can be used to screen any gene in a large population for single nucleotide substitutions, as well as small deletions and insertions. Subjects that are either homozygous or heterozygous for a particular allele can both be identified using DHPLC. The advantage of DHPLC is that it enables the rapid, sensitive, accurate and inexpensive identification of polymorphisms and mutations in an automated fashion. Of greatest importance for this project is the evidence that DHPLC possesses a sensitivity and specificity for mutation detection approaching 100% (Liu, Smith et al. 1998; O'Donovan, Oefner et al. 1998; Arnold, Gross et al. 1999; Choy, Dabora et al. 1999; Gross, Arnold et al. 1999; Jones, Austin et al. 1999; Wagner, Stoppa-Lyonnet et al. 1999; Nickerson, Weirich et al. 2000; Taniguchi, Krishnadath et al. 2000) and that this approach possesses greater sensitivity than gel-based assays.

The sensitivity and accuracy of DHPLC for detection of genetic alterations was probably best demonstrated by a quality control study (Bernstein, Teraoka et al. 2003) performed by the WECARE (Women's Environment, Cancer and Radiation Epidemiology) Study Collaborative Group. There are four international laboratory centers (including the laboratory of Dr. Rosenstein, a co-investigator in this project) that are in the process of screening more than 2000 breast cancer patients for mutations and polymorphisms in a variety of genes associated with DNA repair and radiation responses. The purpose of this quality control study was to investigate the sensitivity and specificity of DHPLC for the detection of ATM mutations and polymorphisms. A panel of 19 DNA samples consisting of 4 unaffected controls, 2 heterozygous carriers, and 13 ataxia telangiectasia patients was supplied in a blinded fashion to each of the four laboratories and screened using DHPLC. Prior screening by Single-Strand Conformation Polymorphism (SSCP) and Protein Truncation Test (PTT) had detected 19 mutations among these samples; 18 of these were detected by DHPLC, an efficiency of 95%. In addition to these 18 mutations, DHPLC screening identified 6 new mutations not detected in prior screening. No mutations were identified in control samples by DHPLC, nor were there excess mutations identified in any ataxia telangiectasia patient or carrier sample, suggesting a low rate of false positives.

#### 10.5 Coding of Samples

Specimens will be given a Study ID number and will be otherwise de-identified for privacy protection. The study data manager will keep the list of samples. Any residual blood specimen after performing the listed laboratory studies will be destroyed.

#### 11 INVESTIGATOR RESOURCES

#### 11.1 Qualifications

Drs. Perez and Huppert and will be responsible for the accrual and care of study patients. Victor Ty will be in charge of study screening, eligibility checklist and will participate in the process of acquisition of an informed consent, after the faculty has discussed the trial with the patient. Victor Ty will also provide the research nursing component of the study, including performing the QOL assessment of the patients.

Drs. Rosenstein and DeWyngaert provide the necessary expertise in radiobiology and physics to conduct the proposed study. Dr. Goldberg will oversee the statistical analyses and collaborate in the interpretation and reporting of the study results. Benjamin Levinson will participate in the ongoing monitoring of this study and statistical analyses.

# 11.2 Use of NYU Facilities

Therapy will be administered in the Department of Radiation Oncology at the Clinical Cancer Center and at Tisch Hospital.

#### 11.3 Conflict of Interest

There are no conflicts of interest to declare.

#### 12 STUDY CALENDAR

| Study Procedure | Pre<br>Treatment | Weekly | Last week | Post Treatment (day 45 - 60) | Post Treatment (once/year) |
|---|---|---|---|---|---|
| History & Physical | X | | | | |
| Mammogram and/or breast MRI <sup>a</sup> | X | | | | Xb |
| Lumpectomy pathology report | X | | | | |
| BREAST-focused exam, KPS | X | X | | X | X |
| Lymphedema assessment | X | | X | | X |
| Blood for TGF-BETA Polymorphisms and other related research studies | X | | Xc | | |
| Quality of Life Questionnaires <sup>d</sup> | X | | X | X | X |
| LENT/SOMA assessment <sup>e</sup> | | | | | X |
| Thyroid Testing (TSH, T <sub>4</sub> ) | X | | | | X |

- a. Standard mammogram or MRI for both breasts.
- b. At each follow-up visit beginning 1 year after completion of radiation treatment a non invasive measurement of fibrosis in the treated breast will be performed using clinical breast exam.
- c. Last day of treatment, after last dose of radiation
- d. QOL will be assessed using the RTOG validated self-assessment questionnaires QLB & QLF (see Appendix 3) at baseline, week 3, day 45 60 and 2-yr follow-ups.
- e. Patients will be seen after completion of treatment at day 45 60 and then yearly for 5 years total follow up to assess long term sequelae by LENT/SOMA scale.

# 13 DATA REPORTING / REGULATORY CONSIDERATIONS

# 13.1 Monitoring Plan

An internal Data and Safety Monitoring Committee (DSMC) of the NYUCI is the monitoring board for this study. The committee will review safety at scheduled intervals (not less than once/year) and at the time of planned interim analyses described in Section 9 according to the NYUCI DSMC Charter.

# 13.2 Stopping Rules (for the individual patient and for the study as a whole)

If safety concerns arise, the DSMC will identify these concerns and recommend modification or termination of the clinical trial. In case of grade 3 acute skin toxicity, the dose per fraction of the remaining treatment fractions will be reduced to 2 Gy/fraction until completion. The clinical trial will be stopped early if regional nodal recurrence is greater than expected (5% of patients) as described in Section 14.

# 13.3 Data Management

Data will be entered into the Oracle Clinical database and maintained at NYUSOM under the direction of staff in the BDM core.

THE ORACLE SYSTEM PROVIDES AUDIT trails that track creation and modification of records that includes userID and time stamp. Once entered, the data are subjected to validation procedures that are executed either immediately or upon saving the eCRF page or during the batch validation process. Validation failures that are identified before the page is saved can be corrected immediately. Validation failures during saving of the eCRF page and during batch validation processes will generate a discrepancy. Depending on the database account privileges, the data managers may be able to correct a discrepancy or if not, route it to the project data manager at NYU who can take appropriate action to correct the problem. Data clarification forms can also be printed out when necessary to be sent to the project data manager. Once the discrepancy is closed, by marking "resolved" or "irresolvable", the data are marked clean and an audit trail is generated by the system.

All key end points will be source verified by a second person and errors will be corrected. Once the data are verified and all discrepancies are closed, the data can be locked/frozen. Locking and freezing can be done at different granular levels and will follow institutional SOPs and any specific requirements for the project.

Security measures that will be taken in order to protect patient data will include firewall technology and database level security which will be achieved by assigning roles and privileges to different levels of users and by requiring that the users authenticate themselves using userID and password. Additional security for data transfer between remote clients and servers will be achieved by using digital certificates/SSL. All data will be backed-up to tape periodically according to the Institutional SOPs. All data will be stored for at least 5 years following the termination of this study.

# 13.4 Confidentiality

The medical, hospital and research records associated with this study are considered confidential. Members of the treating team and designated study assistants will have access to the records as required to administer treatment and comply with the protocol. Neither the name nor any other identifying information for an individual will be used for reporting or publication regarding this study. All laboratory and baseline data will be de-identified and transferred via

secure links to the BDM core at NYU School of Medicine. Patient records will be made available for inspection to auditing agencies to satisfy regulatory requirements.

#### 14 STATISTICAL CONSIDERATIONS

# 14.1 Endpoints/Objectives:

The primary objectives of this study are to:

- 1. To evaluate feasibility of prone IMRT to breast, level I- III (includes Cohort A) and supraclavicular nodes (physics and dosimetry parameters).
- 2. To estimate acute toxicity of prone IMRT to breast, level I- III (includes Cohort A) and supraclavicular nodes

# Secondary objectives are to:

- 1. estimate the incidence of re-simulation to improve dosimetry after initial prone set-up
- 2. evaluate changes in QOL of patients assessed at baseline and after treatment
- 3. estimate incidence of late radiation toxicity (e.g., lymphedema, fibrosis and telangiectasia) and to examine genetic determinants of breast fibrosis

#### Exploratory objectives include:

Estimation of local recurrence rates; estimation of median disease-free survival; estimation of median time to progression, and estimation of median overall survival time.

- 14.2 Statistical Considerations, Sample Size and Interim Analysis Plans
- 14.3 Statistical Analysis

Descriptive statistics will be provided for all demographic and disease characteristics of patients at baseline using frequency distributions for qualitative variables and summary statistics (e.g., median, mean, etc.) and graphical displays (e.g., boxplots) for quantitative variables.

# 14.3.1 Primary Endpoints

The primary outcome of this study is the proportion of patients with acute toxicity greater than grade 2 (Skin toxicities grade 3 and above) occurring within 60 days after first day of treatment. This rate will be estimated with an exact 95% confidence interval. Treatment feasibility will be evaluated for each patient by the ability to meet all physics dose constraints as outlined in section 7.5.6. The proportion of patients who meet the constraints will be estimated with an exact 95% confidence interval.


#### 14.4 Accrual estimates

Estimated number of eligible patients for this trial is 4 - 6 patients per month. Since the recent publication of Giuliano AE (JAMA, 2011 Feb 9; 305(6):606-70), fewer axillary node dissection are being performed nationwide. Consequently, it is expected that the accrual to study NYU 09-0623 may slow down, because of fewer eligible patients. We expect to accrue 104 patients over 5 years.

#### 14.5 Sample Size Considerations/Interim Analysis

The primary endpoint for the estimation of sample size is the proportion of patients with acute skin toxicity of greater than grade 2 occurring within 60 days after first day of treatment. Overall, the regimen will be considered to be unacceptable if more than 5% of patients have acute skin toxicity of greater than grade 2. With 104 patients enrolled in this study, we will have 80% power at a two-sided overall alpha level of 0.05 to test the null hypothesis that the proportion of patients with acute skin toxicity of greater than grade 2 is 0.05. With one interim analysis when 52 patients are evaluable for acute skin toxicity, Table 9 below provides the stopping boundaries for the alternative hypothesis that this proportion is greater than 0.10.

Table 9 - Stopping Boundaries for the Proportion of Patients with Acute Skin Toxicity > Grade 2 based on Pocock Boundaries, Overall 2-sided  $\alpha = 0.05$ , Power =80%. H<sub>0</sub>=0.05; H<sub>1</sub>=0.10 [calculations from EAST 5.2, Cytel, 2008].

| Analysis | Number of | Reject H <sub>0</sub> =0.05 | Reject H <sub>0</sub> =0.05 | Reject H <sub>0</sub> =0.05 |
|---|---|---|---|---|
| | Patients | | | |
| | | Proportion observed | z-statistic | p-value |
| Interim | <mark>52</mark> | ≥ 0.1153 | ≥ 2.57 | ≤ 0.031 |
| Final | 104 | ≥ 0.097 | ≥ 2.201 | ≤ 0.028 |

Additional monitoring will be carried out to estimate the proportion of patients with > grade 2 lymphedema. To test the null hypothesis that this proportion is 0.10 against the alternative that the proportion is 0.19, with 2-sided overall alpha level of 0.05 and power of 78%, at the time of the first interim analysis for skin toxicity, we can reject the null hypothesis if the observed proportion is  $\geq$ 0.19; at the final analysis, we can reject the null hypothesis if the observed proportion is  $\geq$ 0.165 based on Pocock boundaries. There is no adjustment for these two parallel analyses.

With 104 patients, we can estimate the exact 95% confidence interval for the proportion of patients for whom this procedure is feasible with a lower limit of 0.89 or greater if the observed proportion of patients is 0.95 or greater [calculations from PASS, NCSS, LLC (2008), J. Hintze, Kaysville, UT].

Safety Stopping Rule; In addition, regional nodal recurrence will be monitored as the study progresses. If we enroll 104 patients over a three year period with follow-up of one year after the last patient is entered, the regimen will be considered ineffective if the null hypothesis that the proportion of regional nodal recurrences is 5% is rejected at an interim review.

Regional nodal recurrence is defined as recurrence within the axilla, level III or supraclavicular nodes, documented by PET-CT imaging and/or biopsy.

With 5 interim looks (every 21 patients who are followed for at least 1 year), with Pocock stopping boundaries, the trial would be stopped if the observed numbers of regional nodal recurrences are greater than or equal to 1 of the first 21 patients, and greater than 2, 4, 6, and 8 respectively at the second – fifth looks with an overall 1-sided alpha level of 0.05 and power of 0.62 [Calculations from EAST 5.2, Cytel, Inc., 2008].

#### REFERENCES

Archambeau, J. O., R. Pezner, et al. (1995). "Pathophysiology of irradiated skin and breast." <u>Int</u> J Radiat Oncol Biol Phys **31**(5): 1171-85.

- Arnold, N., E. Gross, et al. (1999). "A highly sensitive, fast, and economical technique for mutation analysis in hereditary breast and ovarian cancers." Hum Mutat 14(4): 333-9.
- Atencio, D. P., C. M. Iannuzzi, et al. (2001). "Screening breast cancer patients for ATM mutations and polymorphisms by using denaturing high-performance liquid chromatography." Environ Mol Mutagen **38**(2-3): 200-8.
- Baillet, F., M. Housset, et al. (1990). "The use of a specific hypofractionated radiation therapy regimen versus classical fractionation in the treatment of breast cancer: a randomized study of 230 patients." Int J Radiat Oncol Biol Phys 19(5): 1131-3.
- Bar Ad, V., A. Cheville, et al. (2009). "Time Course of Mild Arm Lymphedema After Breast Conservation Treatment for Early-Stage Breast Cancer." Int J Radiat Oncol Biol Phys.
- Barendsen, G. W. (1982). "Dose fractionation, dose rate and iso-effect relationships for normal tissue responses." <u>Int J Radiat Oncol Biol Phys</u> **8**(11): 1981-97.
- Bartelink, H., J. C. Horiot, et al. (2001). "Recurrence rates after treatment of breast cancer with standard radiotherapy with or without additional radiation." N Engl J Med 345(19): 1378-87.
- Bartelink, H., J. C. Horiot, et al. (2007). "Impact of a higher radiation dose on local control and survival in breast-conserving therapy of early breast cancer: 10-year results of the randomized boost versus no boost EORTC 22881-10882 trial." <u>J Clin Oncol</u> 25(22): 3259-65.
- Bernstein, J. L., S. Teraoka, et al. (2003). "Designing and implementing quality control for multi-center screening of mutations in the ATM gene among women with breast cancer." Hum Mutat 21(5): 542-50.
- Chang, D. T., S. J. Feigenberg, et al. (2007). "Long-term outcomes in breast cancer patients with ten or more positive axillary nodes treated with combined-modality therapy: the importance of radiation field selection." Int J Radiat Oncol Biol Phys 67(4): 1043-51.
- Choy, Y. S., S. L. Dabora, et al. (1999). "Superiority of denaturing high performance liquid chromatography over single-stranded conformation and conformation-sensitive gel electrophoresis for mutation detection in TSC2." <u>Ann Hum Genet</u> **63** ( **Pt 5**): 383-91.
- Darby, S. C., P. McGale, et al. (2005). "Long-term mortality from heart disease and lung cancer after radiotherapy for early breast cancer: prospective cohort study of about 300,000 women in US SEER cancer registries." <u>Lancet Oncol</u> **6**(8): 557-65.
- Deutsch, M., S. Land, et al. (2008). "The incidence of arm edema in women with breast cancer randomized on the National Surgical Adjuvant Breast and Bowel Project study B-04 to radical mastectomy versus total mastectomy and radiotherapy versus total mastectomy alone." Int J Radiat Oncol Biol Phys **70**(4): 1020-4.
- Donegan, W. L., S. B. Stine, et al. (1993). "Implications of extracapsular nodal metastases for treatment and prognosis of breast cancer." <u>Cancer</u> **72**(3): 778-82.
- Douglas, B. G. and J. F. Fowler (1976). "The effect of multiple small doses of x rays on skin reactions in the mouse and a basic interpretation." Radiat Res **66**(2): 401-26.

Fisher, B., S. Anderson, et al. (2002). "Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer." N Engl J Med 347(16): 1233-41.

- Formenti, S. C. (2005). "External-beam partial-breast irradiation." <u>Semin Radiat Oncol</u> **15**(2): 92-9.
- Formenti, S. C., D. Gidea-Addeo, et al. (2007). "Phase I-II trial of prone accelerated intensity modulated radiation therapy to the breast to optimally spare normal tissue." <u>J Clin Oncol</u> **25**(16): 2236-42.
- Fowler, J. (1989). "The linear-quadratic formula and progress in fractionated radiotherapy." <u>Br J</u> Radiol **62**: 679-694.
- Garg, A. K., E. A. Strom, et al. (2004). "T3 disease at presentation or pathologic involvement of four or more lymph nodes predict for locoregional recurrence in stage II breast cancer treated with neoadjuvant chemotherapy and mastectomy without radiotherapy." <u>Int J Radiat Oncol Biol Phys</u> **59**(1): 138-45.
- Gross, E., N. Arnold, et al. (1999). "A comparison of BRCA1 mutation analysis by direct sequencing, SSCP and DHPLC." <u>Hum Genet</u> **105**(1-2): 72-8.
- Harris, E. E., W. T. Hwang, et al. (2003). "Prognosis after regional lymph node recurrence in patients with stage I-II breast carcinoma treated with breast conservation therapy." <u>Cancer</u> **98**(10): 2144-51.
- Haustermans, K., J. Fowler, et al. (1998). "Relationship between potential doubling time (Tpot), labeling index and duration of DNA synthesis in 60 esophageal and 35 breast tumors: Is it worthwhile to measure Tpot?" Radiother Oncol **46**(2): 157-67.
- Hayes, S. B., G. M. Freedman, et al. (2008). "Does axillary boost increase lymphedema compared with supraclavicular radiation alone after breast conservation?" Int J Radiat Oncol Biol Phys **72**(5): 1449-55.
- Hoeller, U., S. Tribius, et al. (2003). "Increasing the rate of late toxicity by changing the score? A comparison of RTOG/EORTC and LENT/SOMA scores." Int J Radiat Oncol Biol Phys **55**(4): 1013-8.
- Huang, E. H., S. L. Tucker, et al. (2005). "Predictors of locoregional recurrence in patients with locally advanced breast cancer treated with neoadjuvant chemotherapy, mastectomy, and radiotherapy." <u>Int J Radiat Oncol Biol Phys</u> **62**(2): 351-7.
- Huber, C. G., P. J. Oefner, et al. (1993). "High-resolution liquid chromatography of oligonucleotides on nonporous alkylated styrene-divinylbenzene copolymers." <u>Anal Biochem</u> **212**(2): 351-8.
- Huber, C. G., P. J. Oefner, et al. (1993). "High-resolution liquid chromatography of DNA fragments on non-porous poly(styrene-divinylbenzene) particles." <u>Nucleic Acids Res</u> **21**(5): 1061-6.
- Iannuzzi, C. M., D. P. Atencio, et al. (2002). "ATM mutations in female breast cancer patients predict for an increase in radiation-induced late effects." <u>Int J Radiat Oncol Biol Phys</u> **52**(3): 606-13.
- James Melissa, L., M. Lehman, et al. (2008) "Fraction size in radiation treatment for breast conservation in early breast cancer." <u>Cochrane Database of Systematic Reviews</u> DOI: 10.1002/14651858.CD003860.pub2.
- Jones, A. C., J. Austin, et al. (1999). "Optimal temperature selection for mutation detection by

- denaturing HPLC and comparison to single-stranded conformation polymorphism and heteroduplex analysis." <u>Clin Chem</u> **45**(8 Pt 1): 1133-40.
- Keramopoulos, A., C. Tsionou, et al. (1993). "Arm morbidity following treatment of breast cancer with total axillary dissection: a multivariated approach." Oncology **50**(6): 445-9.
- Kuklin, A., K. Munson, et al. (1997). "Detection of single-nucleotide polymorphisms with the WAVE DNA fragment analysis system." Genet Test 1(3): 201-6.
- Kurtz, J. M. (2005). "The clinical radiobiology of breast cancer radiotherapy." <u>Radiother Oncol</u> **75**(1): 6-8.
- Lea, D. (1942). "The mechanism of the induction by radiation of chromosome aberrations." <u>J</u> <u>Genet</u> **44**(13): 216-245.
- Liengsawangwong, R., T. K. Yu, et al. (2007). "Treatment optimization using computed tomography-delineated targets should be used for supraclavicular irradiation for breast cancer." <u>Int J Radiat Oncol Biol Phys</u> **69**(3): 711-5.
- Liu, W., D. I. Smith, et al. (1998). "Denaturing high performance liquid chromatography (DHPLC) used in the detection of germline and somatic mutations." <u>Nucleic Acids Res</u> **26**(6): 1396-400.
- Lukens, J. N., N. Vapiwala, et al. (2009). "Regional nodal recurrence after breast conservation treatment with radiotherapy for women with early-stage breast carcinoma." <u>Int J Radiat Oncol Biol Phys</u> **73**(5): 1475-81.
- Matthews, J., B. Meeker, et al. (1989). "Response of human tumor cell lines in vitro to fractionated irradiation." Int J Radiat Oncol Biol Phys **16**: 133-138.
- Moran, M. S. and B. G. Haffty (2002). "Local-regional breast cancer recurrence: prognostic groups based on patterns of failure." <u>Breast J</u> 8(2): 81-7.
- Nickerson, M. L., G. Weirich, et al. (2000). "Signature-based analysis of MET proto-oncogene mutations using DHPLC." <u>Hum Mutat</u> **16**(1): 68-76.
- O'Donovan, M. C., P. J. Oefner, et al. (1998). "Blind analysis of denaturing high-performance liquid chromatography as a tool for mutation detection." Genomics **52**(1): 44-9.
- Oefner, P. J. and P. A. Underhill (1998). DNA mutation detection using denaturing high performance liquid chromatography (DHPLC). <u>Current protocols in Human Genetics</u>. **7.10.1-7.10.12**.
- Powell, S., J. Cooke, et al. (1990). "Radiation-induced brachial plexus injury: follow-up of two different fractionation schedules." <u>Radiother Oncol</u> **18**(3): 213-20.
- Quarmby, S., H. Fakhoury, et al. (2003). "Association of transforming growth factor beta-1 single nucleotide polymorphisms with radiation-induced damage to normal tissues in breast cancer patients." <u>Int J Radiat Biol</u> **79**(2): 137-43.
- Reinertsen, K. V., M. Cvancarova, et al. (2009). "Thyroid Function in Women after Multimodal Treatment for Breast Cancer Stage II/III: Comparison with Controls from a Population Sample." Int J Radiat Oncol Biol Phys.
- Shelbourne, C. D. (1992). <u>Measuring functioning and well-being: the medical outcomes study approach</u>. Durham, Duke University Press.
- Stanton, A. L., L. Krishnan, et al. (2001). "Form or function? Part 1. Subjective cosmetic and functional correlates of quality of life in women treated with breast-conserving surgical procedures and radiotherapy." <u>Cancer</u> **91**(12): 2273-81.
- Stanton, P. D., T. G. Cooke, et al. (1996). "Cell kinetics in vivo of human breast cancer." Br J

- <u>Surg</u> **83**(1): 98-102.
- Steel, G., J. Deacon, et al. (1987). "The dose-rate effect in human tumour cells." <u>Radiother</u> Oncol **9**: 299-310.
- Taghian, A., J. H. Jeong, et al. (2004). "Patterns of locoregional failure in patients with operable breast cancer treated by mastectomy and adjuvant chemotherapy with or without tamoxifen and without radiotherapy: results from five National Surgical Adjuvant Breast and Bowel Project randomized clinical trials." <u>J Clin Oncol</u> 22(21): 4247-54.
- Taniguchi, K., K. Krishnadath, et al. (2000). <u>High sensitivity of denaturing high performance liquid chromatography (DHPLC) in detection of p53 mutations in adenocarcinoma of the esophagus</u>. Proceedings of the 91st Annual Meeting of the American Association for Cancer Research.
- Thames, H., S. Bentzen, et al. (1990). "Time-dose factors in radiotherapy: A review of the human data." Radiother Oncol **19**(219-235).
- Thames, H. and J. Hendry (1987). <u>Fractionation in Radiotherapy</u>. London New York, Taylor and Francis.
- Tian, L., Z. Jun, et al. (2008). <u>Measurements of Radiation-Induced Skin Changes in Breast-Cancer Radiation Therapy Using Ultrasonic Imaging</u>. BioMedical Engineering and Informatics, 2008. BMEI 2008. International Conference on.
- Travis, E. and S. Tucker (1987). "Isoeffect models and fractionated radiation therapy." <u>Int J Radiat Oncol Biol Phys</u> **13**: 283-287.
- Turesson, I. and H. Thames (1989). "Repair capacity and kinetics of human skin during fractionated radiotherapy: Erythema. Desquamation, and telangiectasia after 3 and 5 years follow-up." Int J Radiat Oncol Biol Phys **15**: 169-188.
- Wagner, T., D. Stoppa-Lyonnet, et al. (1999). "Denaturing high-performance liquid chromatography detects reliably BRCA1 and BRCA2 mutations." <u>Genomics</u> **62**(3): 369-76.
- Ware, J. E., Jr. and C. D. Sherbourne (1992). "The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection." Med Care 30(6): 473-83.
- Whelan, T., R. MacKenzie, et al. (2002). "Randomized trial of breast irradiation schedules after lumpectomy for women with lymph node-negative breast cancer." <u>J Natl Cancer Inst</u> **94**(15): 1143-50.
- Williams, M., J. Denekamp, et al. (1985). "A review of / ratios for experimental tumors: Implications for clinical studies of altered fractionation." Int J Radiat Oncol Biol Phys 11: 87-96
- Yamada, Y., I. Ackerman, et al. (1999). "Does the dose fractionation schedule influence local control of adjuvant radiotherapy for early stage breast cancer?" <u>Int J Radiat Oncol Biol Phys</u> **44**: 99-104.

### **APPENDICIES**

## APPENDIX 1 – COMMON TOXICITY CRITERIA

Acute Toxicity from Common Terminology Criteria for Adverse Events v3.0 (CTCAE), Published: August 9, 2006

| | Grade 0 Grade 1 | | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|---|
| FATIGUE | Faint erythema or dry | | Moderate or causing difficulty performing some ADL | culty performing some | |
| RADIATION DERMATITIS | | | Moderate to brisk<br>erythema; patchy moist<br>desquamation, mostly<br>confined to skin folds and<br>creases; moderate edema | Moist desquamation<br>other than skin folds and<br>creases; bleeding induced<br>by minor trauma<br>or abrasion | Skin necrosis or<br>ulceration of full<br>thickness dermis;<br>spontaneous bleeding<br>from involved site |
| PAIN No pain | | Mild pain not<br>Interfering<br>with function | Moderate pain; pain or<br>analgesics interfering with<br>function, but<br>not interfering with ADL | Severe pain; pain or<br>analgesics severely<br>interfering with ADL | Disabling |

| Table 1. RTOG/EORTC and LENT/SOMA classification of late effects | | | | |
|---|---|---|---|---|
| RTOG/EORTC | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Skin | Slight atrophy, pigmentation change, some hair loss | Patchy atrophy, moderate<br>telangiectasia, total<br>hair loss | Marked atrophy, gross telangiectasia | Ulceration |
| Subcutaneous tissue | Slight induration (fibrosis),<br>and loss of subcutaneous<br>fat | Moderate fibrosis, but<br>asymptomatic; slight<br>field contracture,<br>≤10% linear reduction | Severe induration and loss<br>of subcutaneous tissue,<br>field contracture, ≥10%<br>linear reduction | Necrosis |
| LENT/SOMA | | =1070 Inical reduction | mich reddenon | |
| Breast | | | | |
| Subjective | | | | |
| Pain | Occasional and minimal<br>Hypersensation, pruritus | Intermittent and tolerable | Persistent and intense | Refractory and<br>excruciating |
| Objective | 21 | | | J |
| Telangiectasia | <1 cm <sup>2</sup> | $1-4 \text{ cm}^2$ | >4 cm <sup>2</sup> | |
| Fibrosis | Barely palpable, increased density | Definite increased<br>intensity and firmness | Very marked density,<br>retraction, and fixation | |
| Edema | Asymptomatic | Symptomatic | Secondary dysfunction | |
| Retraction, atrophy | 10-25% | >25-40% | >40-75% | Whole breast |
| Ulcer | Epidermal only, <1 cm <sup>2</sup> | Dermal only, >1 cm <sup>2</sup> | Subcutaneous | Bone exposed,<br>necrosis |
| Lymphedema, arm<br>circumference | 2-4-cm increase | >4-6-cm increase | >6-cm increase | Useless arm |
| Skin<br>Pigmentation change | Transitory, slight | Permanent, marked | _ | _ |

Abbreviations: RTOG = Radiation Therapy Oncology Group; EORTC = European Organization for Research and Treatment of Cancer; LENT = Late Effects Normal Tissue Task Force; SOMA = subjective, objective, management, and analytic.

## **APPENDIX 2 – TOXICITY TRACKING FORM**



Department of Radiation Oncology NYU Hospitals Center 550 First Avenue New York, NY 10016

#### PHYSICIAN'S PROGRESS NOTE

| Progress note: | 7/ | or evaluation and pro | gress of treatment (see | notes below) | |
|---|---|---|---|---|---|
| - Togress note | | | W W | 76 Va 97 X 36 M | |
| - | | | | | |
| ======================================= | | | | | |
| - | | | | | |
| - | | | | | |
| Please indicate 1 | Grade 0 | o Radiation Treatment Grade 1 | on the following chart: Grade 2 | Grade 3 | Grade 4 |
| FATIGUE | No change | Mild fatigue over<br>baseline | Moderate or causing<br>difficulty performing<br>some ADL | Severe fatigue interfering<br>with ADL | Disabling |
| DIATION DERMATITIS | No change | Faint erythema or dry<br>desquamation | Moderate to brisk<br>erythema; patchy moist<br>desquamation, mostly<br>confined to skin folds and<br>creases; moderate edema | Moist desquamation other than skin folds and creases; bleeding induced by minor trauma or abrasion | Skin necrosis or<br>ulceration of full<br>thickness dermis;<br>spontaneous bleeding<br>from involved site |
| DIATION DERMATITIS | | | erythema; patchy moist<br>desquamation, mostly<br>confined to skin folds and | other than skin folds and<br>creases; bleeding induced<br>by minor trauma | ulceration of full<br>thickness dermis;<br>spontaneous bleeding |

## APPENDIX 3 – QUALITY OF LIFE QUESTIONNAIRES

| Accele | -0623 Phase I-II Study of Prone<br>erated Breast and Nodal IMRT<br>of Life Questionnaire - Baseline | Form QLB (01-25-2005)<br> |
|---|---|---|
| Patient Initials , First Middle | Patient<br>Study ID | |
| Participants should complete this questionn a clinical staff member. Fill in the items list through 7 and give the questionnaire to the questionnaire, verify that the date has been Please administer the questionnaire at an of the patient, then call to ask for the patient's questionnaire fail, a B-39 QMD form should be the patient of the patient. | ed on this page, print the patient's study patient for completion. After the patient recorded at the top of page 2. Office visit if possible. If that is not possion responses over the phone. If all efforts | ID at the top of pages 2<br>t has completed the<br>ble, mail the questionnaire to |
| | Mark Circles Like This: → ● | |
| Institution Name / Affiliate Name Staff Member Administering Form | | |
| Last Name 171 Are data amended? OYes (If yes, circ | First Name | Phone |
| Time point for this questionnaire (I Baseline (after consent) | Do not mark in this box.) | |
| CONTROL OF THE PROPERTY OF THE | s being filled out: (Mark one.) | th narticinant |
| O By participant in doctor's office O By participant not in doctor's office | O By clinical staff, on phone wi<br>O Other | тп раптісірапт |

Record the participant's study ID on each of the remaining pages before giving the questionnaire to the participant.



Version 03/23/2017 NYU 09-0623

| •••• | Form QLB (01-25-2005)<br> |
|---|---|
| | Patient<br>Study ID |
| Date this questionnaire is completed: | Day Year |
| (For example, if you were completing the questi- | onnaire on September 8, 2004, you would |

write 09 08 2004 in the boxes.)

Thank you for completing this questionnaire.

We are interested in your evaluation of your physical appearance and functioning since you have been treated for breast cancer. Please rate the following items on this four-point scale, according to your evaluation at this point in time

#### Difference between treated and untreated breast and area None Slight Moderate Large 3 1 Breast size 2 Breast texture (hardening) 2 3 2 3 Arm heaviness 2 3 4 Nipple appearance 4 2 5 Shoulder movement 6 Arm movement 2 7 Breast pain 8 Ability to lift objects 2 2 9 Fit of shirt sleeve 10 Breast tenderness 2 2 11 Shoulder stiffness 2 12 Breast shape 13 Breast elevation (how high the breast is) 2 2 14 Scar tissue 2 15 Shoulder pain 2 16 Arm pain 17 Arm swelling 18 Breast swelling 2 19 Arm stiffness 2 2 20 Fit of bra 2 21 Breast sensitivity 1 22 Fit of clothing 2

| | **** | | | | | | | Fo | rm QLB (01<br>Pa | -25-2005)<br>age 3 of 7 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Patie<br>Stud | 1735/T | | | |
| Ple<br>pt | are interested<br>ase answer the<br>ions are labele<br>ile as appropria | following d at the e | g question<br>nd-points | ns by <u>circ</u><br>sonly. H | ding one (<br>owever, y | 1) numbe | er. Pleas | e note th | at the res | sponse |
| ١. | To what extent | has your | surgery | disrupte | <b>d</b> your no | rmal <u>dail</u> | y activitie | <u>s</u> ? | | |
| | 0 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| 2. | Not at all<br>To what extent | t has your | surgery | disrupte | <b>d</b> your no | rmal <u>recr</u> | eational | activities | ? | A lot |
| | 0 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| 3. | Not at all<br>To what extent<br>friends? | t has your | surgery | disrupte | <b>d</b> your no | rmal <u>acti</u> | vities with | n your far | nily and | A lot |
| | 0 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not at all<br>To what extent | t has your | surgery | disrupte | <b>d</b> your no | rmal <u>slee</u> | p pattern | <u>ı</u> ? | | A lot |
| | 0 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not at all<br>To what extent | t has your | surgery | reduced | your <u>enj</u> o | yment of | life? | | | A lot |
| | 0 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| i. | Not at all<br>To what extent<br>time off, not ge<br>pay, please ch | etting don | e as muc | h as you' | | f you do i | not work | | | |
| | 0 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not at all<br>How satisfied | are you v | vith the <u>le</u> | ength of t | ime your | treatment | : has take | n to this | point in t | A lot<br>ime? |
| | 0 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not at all<br>How <b>disruptiv</b><br>and close frien | | ır surgery | been to | the <u>other</u> | importan | it people | in your li | <u>fe</u> (e.g., f | A lot<br>amily |
| | 0 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | Not at all | | 82 55 | | | | | | | A lot |

| | | | | | | | | | | | For | m QLB (01-25-20<br>Page 4 c | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Patient<br>Study ID | | | | Τ |
| wee | | each c | | | | | | | | | | the past 4<br>vay you have | ; |
| Ηον | w much of | f the t | ime <u>dur</u> | ing the | past 4 | weeks | <u>§</u> | | | | | | |
| | | | | | | All<br>of the<br>time | of | ost<br>the<br>ne | Some of the time | | A little<br>of the<br>time | None<br>of the<br>time | |
| 1. | Did you fe | el full | of life? | ,<br> | | 1 | : | 2 | 3 | | 4 | 5 | |
| 2. | Did you h | ave a | lot of e | nergy? | , | 1 | : | 2 | 3 | | 4 | 5 | |
| 3 | Did you fe | el wo | rn out? | | | 1 | : | 2 | 3 | | 4 | 5 | |
| 4. | Did you fe | el tire | ed? | | | . 1 | ; | 2 | 3 | | 4 | 5 | |
| | Rate you 0 No pain | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10<br>Pain as b<br>can imag | pad as you<br>ine | |
| 6. | Rate you | 12 | | | | | | | | | 51 | 1 | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | |
| | No pain | | | | | | | | | | Pain as b | ad as you<br>ine | |
| 7. | Rate you | r pain | on <u>ave</u> | <u>rage</u> ir | the pa | st four | weeks | (Circ | le one nu | ımb | er.) | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | |
| | No pain | n sessiones | | | | | <b>(0</b> !1- | | | | Pain as b<br>can imag | ad as you<br>ine | |
| 8. | Rate how | | 67707 | 15375 | | | | 550 | (5.0) | _ | 40 | ĺ | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | |
| 0 | No pain | rro.m | the room | ivina t | rootmo | nto or t | okina m | odiool | tions for y | (O.U.III | can imag | ad as you<br>ine | |
| <b>9</b> . | Are you o | | | | eaime | iils Or I | акінд П | ieuicai | uons ior ) | our | раш? | | |

1-4: SF - 36 v2 Vitality and 5-9: BPI Copyright 1991 Charles S. Cleeland, Ph.D. Pain Research Group Used by permission.

| Form QLB | (01-25-200 | (5) |
|----------|------------|-----|
| | Page 5 of | 7 |

| Patient<br>Study ID |
|---------------------|
|---------------------|

By circling one (1) number per line, please indicate how much you have been bothered by each of the following problems in the past four weeks.

| | Not<br>bothered<br>at all | A little<br>bit<br>bothered | Some-<br>what<br>bothered | Bothered<br>quite<br>a bit | Bothered<br>very<br>much |
|---|---|---|---|---|---|
| Fever or shivering (shaking, chills) | 0 | 1 | 22 | 3 | 4 |
| Swelling of breast (breast feels larger) | 0 | 1 | 22 | 3 | 4 |
| Breast heaviness | 0 | 1 | 2 | 3 | 4 |
| Breast warm to touch | 0 | 1 | 2 | 3 | 4 |
| Breast skin is red | 0 | 1 | 2 | 3 | 4 |
| Breast skin is tanned | 0 | 1 | 2 | 3 | 4 |
| Breast skin or area around nipple is pale in color | 0 | 1 | 22 | 3 | 4 |
| Breast skin is flaking or peeling | 0 | 11 | 2 | 3 | 4 |
| Bleeding or fluid leakage from breast | 0 | 1 | 2 | 3 | 4 |
| Breast itching | 0 | 1 | 2 | 3 | 4 |
| Blisters on the breast (or breast skin moist and raw) | 0 | 1 | 2 | 3 | 4 |
| Coughing | 0 | 11 | 2 | 3 | 4 |
| Difficulty breathing | 0 | 1 | 2 | 3 | 4 |
| Muscle aches | 0 | 1 | 2 | 3 | 4 |
| Rib or chest wall pain | 0 | 1 | 2 | 3 | 4 |
| Infections | 0 | 1 | 2 | 3 | 4 |
| Slow healing of breast wounds | 0 | 1 | 2 | 3 | 4 |
| Visible small blood vessels (spider veins) | 0 | 1 | 2 | 3 | 4 |
| Pockmarks or puncture wounds on breast | 0 | 11 | 2 | 3 | 4 |
| Thickening of breast skin | 0 | 1 | 2 | 3 | 4 |
| Hardening of breast | 0 | 1 | 2 | 3 | 4 |
| Breast or nipple numbness | 0 | 1 | 2 | 3 | 4 |
| Sharp shooting pains or twinges in the breast | 0 | 1 | 2 | 3 | 4 |

SCL





| | cling one (1) number per line, pleas<br>If the following problems <u>in the pa</u> | | | ou have b | een both | ered by |
|---|---|---|---|---|---|---|
| | | Not<br>bothered<br>at all | | Some-<br>what<br>bothered | Bothered<br>quite<br>a bit | Bothered<br>very<br>much |
| Bre | east aches | 0 | 1 | 2 | 3 | 4 |
| Bre | east tenderness | 0 | 1 | | | 4 |
| Dec | crease or lack of arousal on breast | 0 | 1 | 2 | 3 | 4 |
| Any | y other problems? (Specify below) | 0 | 1 | 2 | 3 | 4 |
| Spe | ecify other problems: | | | | | |
| nion d | concerning the appearance of your bat best describes how your breast loc EXCELLENT: when compared to | oks <u>now</u> . the untreated | breast or t | he original | appearan | ce of the |
| nion o | EXCELLENT: when compared to breast, there is minimal or no diffe way the breast feels (its texture) is thickening, scar tissue or fluid according to the scar tissue or fluid according | the untreated<br>rence in the si<br>the same or s | breast or t<br>ze or shap<br>slightly diffe | the original<br>e of the tre<br>erent. The | appearan<br>ated brea<br>re may be | ce of the<br>st. The |
| nion o | EXCELLENT: when compared to breast, there is minimal or no diffe way the breast feels (its texture) is thickening, scar tissue or fluid accuthe appearance. GOOD: there is a slight difference compared to the opposite breast of may be some mild reddening or day. | the untreated rence in the sist the same or sumulation with the size or or the original aarkening of the | breast or t<br>ze or shap<br>slightly diffe<br>in the brea<br>shape of t<br>appearance<br>breast. Th | the original<br>e of the tree<br>erent. The<br>est, but not<br>the treated<br>e of the tree<br>ne thickenii | appearan eated brea re may be enough to breast as ated breas | ce of the st. The change |
| nion ord tha | EXCELLENT: when compared to breast, there is minimal or no diffe way the breast feels (its texture) is thickening, scar tissue or fluid accepte appearance. GOOD: there is a slight difference compared to the opposite breast of may be some mild reddening or day within the breast causes only a mile. | the untreated rence in the sist the same or sumulation with the size or or the original arkening of the ld change in the | breast or the present of the present | the original<br>e of the tree<br>erent. The<br>est, but not<br>the treated<br>e of the tree<br>ne thickening | appearan<br>eated brea<br>re may be<br>enough to<br>breast as<br>ated breas<br>ng or scar | ce of the<br>st. The<br>change<br>st. There<br>tissue |
| rd tha | EXCELLENT: when compared to breast, there is minimal or no diffe way the breast feels (its texture) is thickening, scar tissue or fluid accuthe appearance. GOOD: there is a slight difference compared to the opposite breast of may be some mild reddening or day. | the untreated rence in the sis the same or sumulation with the original arkening of the ld change in the size and shape reast. There c | breast or the present of the present | the original<br>e of the tree<br>erent. The<br>est, but not<br>the treated<br>e of the tree<br>ne thickening<br>r size.<br>ated breas<br>lerate thicken | appearant atted breast as atted breast as atted breast ang or scar | ce of the st. The change st. There tissue |
| nion ord tha | EXCELLENT: when compared to breast, there is minimal or no diffe way the breast feels (its texture) is thickening, scar tissue or fluid accepte appearance. GOOD: there is a slight difference compared to the opposite breast or may be some mild reddening or day within the breast causes only a mild FAIR: obvious differences in the sinvolves a quarter or less of the breast local services. | the untreated rence in the sist the same or sumulation with the in the size or or the original arkening of the ld change in the size and shape reast. There coere may be obpearance of the kin changes muscarring and the size and the size and shape reast. | breast or to ze or shape of to appearance breast. The shape of the tree an be modulous color of the tree and be treated by any be obvinickening of the shape of the tree and the shape of t | the original e of the treated e of the treated e of the treated e thickening r size. ated breas lerate thick r changes. oreast involus and de | appearantiated breaster may be enough to breast as ated breasted breasted breasted breasted breasted breasted breasted breaster from more etract from | ce of the st. The change st. There tissue ange scar tissue than a the |
| nion derd that | EXCELLENT: when compared to breast, there is minimal or no diffe way the breast feels (its texture) is thickening, scar tissue or fluid acceptate appearance. GOOD: there is a slight difference compared to the opposite breast or may be some mild reddening or day within the breast causes only a mild FAIR: obvious differences in the sinvolves a quarter or less of the broof the skin and the breast, and the POOR: marked change in the appearance of the breast. Severe | the untreated rence in the sist the same or sumulation with the in the size or or the original arkening of the ld change in the size and shape reast. There core may be observed to the changes must be considered to the changes must be four scarring and the st, may be four | breast or to ze or shape of to appearance breast. The shape of the tree an be modified by the color of the tree and be modified by the color of the tree and be modified by the color of the tree and be obvious color of the tree and be obvious color of the tree and the color of the color of t | the original e of the tree erent. The erent. The erent ist, but not the treated e of the tree ene thickening r size. ated breas lerate thicker changes. It involves and dept the breas erent involves erent | appearantiated breaster may be enough to breast as ated breast as ated breasted breasted breaster in this characterist. This characterist may be breaster from st, which contact from the st. | ce of the st. The change st. There tissue ange scar tissue than a the clearly |
| anion of the rd that 1 2 My satis | EXCELLENT: when compared to breast, there is minimal or no diffe way the breast feels (its texture) is thickening, scar tissue or fluid acceptate appearance. GOOD: there is a slight difference compared to the opposite breast of may be some mild reddening or day within the breast causes only a mild FAIR: obvious differences in the sinvolves a quarter or less of the boof the skin and the breast, and the POOR: marked change in the appearance of the breast. Severe alters the appearance of the breast satisfaction about the treatment and | the untreated rence in the sist the same or sumulation with the in the size or or the original arkening of the ld change in the size and shape reast. There core may be observed to the changes must be considered to the changes must be four scarring and the st, may be four | breast or to ze or shape of to shape of to shape of the tree and be mode of the tree and tree and tr | the original e of the tree erent. The erent. The erent ist, but not the treated e of the tree ene thickening r size. ated breas lerate thicker changes. It involves and dept the breas erent involves erent | appearantiated breaster may be enough to breast as ated breast as ated breasted breasted breaster in this characterist. This characterist may be breaster from st, which contact from the st. | ce of the st. The change st. There tissue ange scar tissue than a the clearly |

| <b>***</b> | | Form QLB (01-25-2005)<br> |
|---|---|---|
| | Patient<br>Study ID | |
| Before any treatment to yo describes your breast size | our breast, the size of your breasts was: (See prior to treatment.) | elect the phrase that best |
| Larger | The same on | Larger |
| on left | both sides | on right |
| The size of your breasts n | now is: (Select the phrase that best describes | s your breast size now.) |
| Larger | The same on | Larger |
| on left | both sides | on right |

Thank you for completing this questionnaire!

RTOG PQ

| | Accelerate | 3 Phase I-II Study o | IMRT | Form QLF(01-25-2005)<br>Page 1 of 6 | |
|---|---|---|---|---|---|
| | Quality of Life | e Questionnaire - F | | | _ |
| Patient , Last First Middle | | | itient<br>udy ID | | |
| Patients who experience complete questionnaires to complete all the quality | after that event. Pati | ients who discontinue | | | |
| The first page is to be conpatient's study ID at the to through 6 and give the quality that | op of pages 2 throug<br>uestionnaire to the p | gh 6 and the assessme<br>atient for completion. | ent time poin<br>After the pat | t at the bottom of pages | |
| Please administer the que<br>questionnaire to the patie<br>administer the scheduled | nt, then call to ask f | or the patient's respon | ses over the | phone. If all efforts to | |
| Institution Name / Affilia | ite Name | | | | |
| Staff Member Administe | ring Form | | | | |
| Last i | Name | First Na | ime | Phone | |
| Are data amended? O | Yes (If yes, circle | the amended items.) | | | |
| | This form is b | peing filled out: (Ma | ark one.) | | _ |
| O By participant in do | ctor's office | O By clinical staff, | on phone | with participant | |
| O By participant not in | n doctor's office | O Other | 12 | | |
| | Mark | Circles Like This: → ● | | | |

assessment time point O End of RT O Day 45-60 O 2 years

Record the assessment time point and participant's Study ID on each of the remaining pages before giving the questionnaire to the participant.

| | | | Form QLF(01-25-2005)<br>Page 2 of 6 |
|---|---|---|---|
| | | Patient<br>Study ID | |
| Date this questionnaire is completed: | Month Day | Year | |

(For example, if you were completing the questionnaire on September 8, 2004, you would write 09 08 2004 in the boxes.)

Thank you for completing this questionnaire.

We are interested in your evaluation of your physical appearance and functioning since you have been treated for breast cancer. Please rate the following items on this four-point scale, according to your evaluation at this point in time.

# Difference between treated and untreated breast and area

| | | Dicast | ana arca | |
|---|---|---|---|---|
| | None | Slight | Moderate | Large |
| 1 Breast size | 1 | 2 | 3 | 4 |
| 2 Breast texture (hardening) | 1 | 2 | 3 | 4 |
| 3 Arm heaviness | 1 | 2 | 3 | 4 |
| 4 Nipple appearance | 1 | 2 | 3 | 4 |
| 5 Shoulder movement | 1 | 2 | 3 | 4 |
| 6 Arm movement | 1 | 2 | 3 | 4 |
| 7 Breast pain | 1 | 2 | 3 | 4 |
| 8 Ability to lift objects | 1 | 2 | 3 | 4 |
| 9 Fit of shirt sleeve | 1 | 2 | 3 | 4 |
| 10 Breast tenderness | 1 | 2 | 3 | 4 |
| 11 Shoulder stiffness | 1 | 2 | 3 | 4 |
| 12 Breast shape | . 1 | 2 | 3 | 4 |
| 13 Breast elevation (how high the breast is) | . 1 | 2 | 3 | 4 |
| 14 Scar tissue | . 1 | 2 | 3 | 4 |
| 15 Shoulder pain | 1 | 2 | 3 | 4 |
| 16 Arm pain | . 1 | 2 | 3 | 4 |
| 17 Arm swelling | 1 | 2 | 3 | 4 |
| 18 Breast swelling | 1 | 2 | 3 | 4 |
| 19 Arm stiffness | 1 | 2 | 3 | 4 |
| 20 Fit of bra | . 1 | 2 | 3 | 4 |
| 21 Breast sensitivity | 1 | 2 | 3 | 4 |
| 22 Fit of clothing | 1 | 2 | 3 | 4 |

| assessment time point | O End of RT | O Day 45-60 | O 2 years | 0 |
|------------------------|---------------|-------------|-----------|---|
| accoconnent time penne | C Lind of Itt | • Du, 10 00 | , | _ |

встоѕ



| | • | | | | | | | | | | Form | QLF(01-2<br>Pag | 5-2005)<br>je 3 of 6 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | Patient<br>Study ID | | | | | T |
| <u>we</u> | | each d | | | | | | | | | you <u>during</u><br>est to the w | | | |
| Ho | w much o | f the t | ime <u>dur</u> | ing the | oast 4 | 1 weeks | | | | | | | | |
| | | | | | ( | All<br>of the<br>time | of | ost<br>the<br>ne | Some<br>of the<br>time | | A little<br>of the<br>time | Nor<br>of t<br>tim | ne | |
| 1. | Did you fe | el ful | l of life? | | | 1 | | 2 | 3 | | 4 | 5 | | |
| 2. | Did you h | ave a | lot of e | nergy? | | 1 | | 2 | 3 | | 4 | 5 | | |
| 3 | Did you fe | el wo | rn out? | | | 1 | : | 2 | 3 | | 4 | 5 | | |
| 4. | Did you fe | el tire | ed? | | | 1 | | 2 | 3 | | 4 | 5 | | |
| 5. | Rate you | r pain | at its <u>w</u><br>2 | <u>rorst</u> in t | he pa | ıst four | weeks. | (Circl | 1 5 | 8 | | | | |
| | | 1 | | <u> </u> | 4 | - J | 0 | 1 | 8 | 9 | 10 | | | |
| | No pain | | | | | | | | | | Pain as b<br>can imagi | | ou | |
| 6. | Rate you | r pain | at its <u>le</u> | ast in th | ne pa | st four v | veeks. | (Circle | e one nur | nbe | er.) | | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | |
| _ | No pain | | | | | | | | | | Pain as b<br>can imagi | | ou | |
| 7. | Rate you | | CMA | ****** | 2000 | 9000 | 4875 | 0.000 | No. | 0.00000 | | | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | |
| | No pain | | | | | | | | | | Pain as b | | ou | |
| 8. | Rate how | v muc | h pain y | ou have | right | t now. ( | Circle | one nu | ımber.) | | | | | |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | |
| | No pain | | | | | | | | | | Pain as b | 150 | ou | |
| 9. | Are you o | | itly rece<br>′es No | | atme | nts or to | aking n | nedicat | tions for y | /ou | r pain? | | | |
| | | | | | | | | | | | | 1 | | |
| | as | sessr | nent tin | ne poin | t 0 | End of R | T O D | ay 45-6 | 0 <b>O</b> 2 ye | ears | 0 | J <sub>┣</sub> | | 1 |
| 1 | -4: SF - 36 v2 | Vitality ar | nd 5-9: BPI | Copyright 1 | 991 Cha | rles S. Clee | land, Ph.D | . Pain Res | search Group | Used | by permission. | | 7 | ] |

Version 03/23/2017 NYU 09-0623

| Form QLF(01-25-20<br>Page 4 |
|-----------------------------|
| Patient<br>Study ID |

By circling one (1) number per line, please indicate how much you have been bothered by each of the following problems <u>in the past four weeks</u>.

| | Not<br>bothered<br>at all | A little<br>bit<br>bothered | Some-<br>what<br>bothered | Bothered<br>quite<br>a bit | Bothered<br>very<br>much |
|---|---|---|---|---|---|
| Fever or shivering (shaking, chills) | 0 | 1 | 2 | 3 | 4 |
| Swelling of breast (breast feels larger) | 0 | 1 | 2 | 3 | 4 |
| Breast heaviness | 0 | 1 | 2 | 3 | 4 |
| Breast warm to touch | 0 | 1 | 2 | 3 | 4 |
| Breast skin is red | 0 | 1 | 2 | 3 | 4 |
| Breast skin is tanned | 0 | 1 | 2 | 3 | 4 |
| Breast skin or area around nipple is pale in color | 0 | 1 | 22 | 3 | 4 |
| Breast skin is flaking or peeling | 0 | 1 | 2 | 3 | 4 |
| Bleeding or fluid leakage from breast | 0 | 1 | 2 | 3 | 4 |
| Breast itching | 0 | 1 | 2 | 3 | 4 |
| Blisters on the breast (or breast skin moist and raw) | 0 | 1 | 22 | 3 | 4 |
| Coughing | 0 | 1 | 2 | 3 | 4 |
| Difficulty breathing | 0 | 1 | 2 | 3 | 4 |
| Muscle aches | 0 | 1 | 2 | 3 | 4 |
| Rib or chest wall pain | 0 | 1 | 2 | 3 | 4 |
| Infections | 0 | 1 | 2 | 3 | 4 |
| Slow healing of breast wounds | 0 | 1 | 2 | 3 | 4 |
| Visible small blood vessels (spider veins) | 0 | 1 | 2 | 3 | 4 |
| Pockmarks or puncture wounds on breast | 0 | 1 | 2 | 3 | 4 |
| Thickening of breast skin | 0 | 1 | 2 | 3 | 4 |
| Hardening of breast | 0 | 1 | 2 | 3 | 4 |
| Breast or nipple numbness | 0 | 1 | 2 | 3 | 4 |
| Sharp shooting pains or twinges in the breast | 0 | 1 | 2 | 3 | 4 |

| assessment time point | O End of RT | O Day 45-60 | O 2 years | 0 |
|-----------------------|-------------|-------------|-----------|---|



| | F | orm | QLF( | 5-200<br>je 5 d |
|---------------|---|-----|------|-----------------|
| Patie<br>Stud | | | | |

By circling one (1) number per line, please indicate how much you have been bothered by each of the following problems in the past four weeks.

| , | Not<br>bothered<br>at all | A little<br>bit<br>bothered | Some-<br>what<br>bothered | Bothered<br>quite<br>a bit | Bothered<br>very<br>much |
|---|---|---|---|---|---|
| Breast aches | 0 | 1 | 2 | 3 | 4 |
| Breast tenderness | 0 | 1 | 22 | 3 | 4 |
| Decrease or lack of arousal on breast | 0 | 1 | 22 | 3 | 4 |
| Tattoos on breast placed for radiation therapy | 0 | 1 | 2 | 3 | 4 |
| Any other problems? (Specify below) | 0 | 1 | 2 | 3 | 4 |

You have been treated with breast conserving therapy for breast cancer. As you know, a reason for choosing this treatment is to keep a breast that looks and feels as close to normal as possible. Your opinion concerning the appearance of your breast is valuable to us. <u>Circle the number</u> next to the word that best describes how your breast looks <u>now</u>.

| 1 | <b>EXCELLENT:</b> when compared to the untreated breast or the original appearance of the breast, there is minimal or no difference in the size or shape of the treated breast. The way the breast feels (its texture) is the same or slightly different. There may be thickening, scar tissue or fluid accumulation within the breast, but not enough to change the appearance. |
|---|---|
| 2 | <b>GOOD:</b> there is a slight difference in the size or shape of the treated breast as compared to the opposite breast or the original appearance of the treated breast. There may be some mild reddening or darkening of the breast. The thickening or scar tissue within the breast causes only a mild change in the shape or size. |
| 3 | <b>FAIR</b> : obvious differences in the size and shape of the treated breast. This change involves a quarter or less of the breast. There can be moderate thickening or scar tissue of the skin and the breast, and there may be obvious color changes. |
| 4 | <b>POOR:</b> marked change in the appearance of the treated breast involving more than a quarter of the breast tissue. The skin changes may be obvious and detract from the appearance of the breast. Severe scarring and thickening of the breast, which clearly alters the appearance of the breast, may be found. |

| assessment time point | O End of RT | O Day 45-60 | O 2 years | 0 |
|-----------------------|-------------|-------------|-----------|---|

SCL and RTOG PQ



| | | | | | Form QLF(01- | -25-2005)<br>age 6 of 6 |
|---|---|---|---|---|---|---|
| | | | | Patient Study ID | | |
| My sat | | ne treatment and | results is: (Selec | ct the phrase tha | t best descri | bes your |
| Totall<br>satisfie | , | mewhat<br>atisfied | Neither<br>satisfied nor<br>dissatisfied | Somewhat<br>dissatisfied | | Totally<br>ssatisfied |
| | | your breast, the | | ısts was: (Selec | t the phrase | that best |
| Large<br>on le | er | | The same on both sides | | | Larger<br>on right |
| The si | ze of your breast | s now is: (Select | the phrase that b | est describes yo | ur breast siz | ze now.) |
| Large<br>on le | | | The same on both sides | | | Larger<br>on right |
| Thank | you for com | pleting this | questionnai | re! | | |
| Γ | assessment tin | ne point O End o | of RT <b>O</b> Day 45-60 | O 2 years O | | |
| RTOG PC | | To the second se | une vender epop 200401€ pp.25-19901 | - Suresquery • suresquery (CES) | | <del>-</del> -7 ■ |



#### NYU 09-0623 Phase I-II Study of Prone Accelerated Breast and Nodal IMRT

| Corm OMD (04 35 3005) |
|-----------------------|
| Form QMD (01-25-2005) |
| Page 1 of 1 |
| Page I OI I |

#### Missing Data Form for Quality of Life Questionnaire

Submit this form whenever a protocol-scheduled Quality of Life (QOL) Questionnaire (i.e., Form QLT, QLP, or QLF) is not filled out by the patient and the assessment cannot be obtained by phone or mail. No missing data form is required for partially completed QOL forms or patients who have died or had a documented breast cancer recurrence or a second primary cancer.

| Patient , | Patient ID |
|---|---|
| Institution Name / Affiliate Name | 1 |
| Person | |
| Completing Form | First Name Phone |
| Today's Date Month Day Year | FIIST NAME FILOTE |
| Are data amended? (check box if yes, and circle amended items) | □Yes |
| Time Point for this | Form (mark one) |
| O Form QLT: Last day of radiation therapy | 0 |
| O Form QLP: 45-60 days after start of radiation therapy | 0 |
| O Form QLF: 2 years after radiation therapy | 0 |
| Reason QOL was Not Assessed<br>During Clinic Visit | Reason QOL was Not Obtained<br>by Phone or Mail |
| (Mark the main reason and add comments below.) | (Mark all that apply and add comments below.) |
| O Staff oversight or understaffing | O Staff oversight or understaffing |
| Staff concerned for patient's medical or emotional condition | O Patient's medical or emotional condition |
| | O Patient refused to complete questionnaire |
| O Patient stated that she was too ill or upset to complete questionnaire | O Staff was unable to contact patient by phone |
| O Patient refused to complete questionnaire for reason other than illness or upset | <ul> <li>Questionnaire was mailed to patient but<br/>she did not return it (for any reason)</li> </ul> |
| O Patient was unavailable (e.g., scheduling or transportation difficulties) | |
| Comments | |

Mark Circles Like This: → ●

